CLINICAL TRIAL: NCT00925002
Title: OPEN-LABEL SAFETY AND EFFICACY EVALUATION OF FX-1006A IN SUBJECTS WITH TRANSTHYRETIN (TTR) AMYLOIDOSIS
Brief Title: Safety And Efficacy Evaluation Of Fx-1006A In Subjects With Transthyretin Amyloidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: FX1A-303; B3461023 (Other: Alias Study Number); 2009-011535-12 (EudraCT Number)
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: ATTR-PN
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label (Active Comparator)
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — 20 mg oral Fx-1006A daily

SUMMARY:
This is a Phase 3, open-label study designed to obtain additional long-term safety and efficacy data for oral tafamidis (20 mg soft gelatin capsule) administered once daily (QD). In addition, this study continued to provide tafamidis to Val30Met subjects who had completed Protocol Fx-006 (a 1-year, open-label extension study to Protocol Fx-005 which was a randomized, double-blind, placebo-controlled, 18-month study to evaluate the safety and efficacy of tafamidis) or non-Val30Met subjects who had completed Protocol Fx1A-201 (a Phase 2, open-label study to evaluate TTR stabilization, safety, and tolerability of tafamidis) for up to 10 years or until subjects had access to tafamidis for ATTR-PN via prescription. Upon regulatory approval for the treatment of ATTR-PN in their respective country and access to prescription tafamidis, subjects may have been withdrawn from the study. Such subjects were considered study completers.

ELIGIBILITY:
Key Inclusion criteria:

* Subject had successfully completed either Protocol Fx-006 or Fx-1A-201.
* Male or female subjects with ATTR-PN who had not undergone liver or heart transplantation at time of enrollment.
* If female, subject was post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control

Key Exclusion criteria:

* Chronic use of non-protocol approved non-steroidal anti-inflammatory drugs (NSAIDs)
* Pregnant or breast feeding female subjects.
* Clinically significant medical condition that, in the opinion of the investigator, would place the subject at an increased risk to participate in the study.
* An alanine aminotransferase (ALT) and aspartate aminotransferase (AST) value >3 × upper limit of normal (ULN) that, in the medical judgment of the investigator, was due to reduced liver function or active liver disease.
* Sexually active males with partners of childbearing potential not using highly effective contraception or not agreeing to continue highly effective contraception for at least 3 months after last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-08-05 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Johns Hopkins Hospital, Baltimore, Maryland, United States
- FLENI, Buenos Aires, Argentina
- Hospital Universitário Clementino Fraga Filho -HUCFF Universidade Federal do Rio de Janeiro, Rio de Jameiro, R.J., Brazil
- Centre d'Investigation Clinique, Créteil, France
- Universitatsklinikum Muenster, Münster, Germany
- Centro per lo Studio e la Cura delle Amiloidosi Sistemiche IRCCS - Policlinico San Matteo, Pavia, Italy
- Portugal (2):
  - Centro Hospitalar Lisboa Norte, EPE- Hospital de Santa Maria, Lisbon
  - Unidade Clinica de Paramiloidose Centro Hospitalar do Porto, EPE - Hospital Geral de Santo António, Porto
- FAP-Teamet Familjar Amyloidos, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Merlini G, Coelho T, Waddington Cruz M, Li H, Stewart M, Ebede B. Evaluation of Mortality During Long-Term Treatment with Tafamidis for Transthyretin Amyloidosis with Polyneuropathy: Clinical Trial Results up to 8.5 Years. Neurol Ther. 2020 Jun;9(1):105-115. doi: 10.1007/s40120-020-00180-w. Epub 2020 Feb 27. PMID 32107748
- [Derived] Huber P, Flynn A, Sultan MB, Li H, Rill D, Ebede B, Gundapaneni B, Schwartz JH. A comprehensive safety profile of tafamidis in patients with transthyretin amyloid polyneuropathy. Amyloid. 2019 Dec;26(4):203-209. doi: 10.1080/13506129.2019.1643714. Epub 2019 Jul 27. PMID 31353964
- [Derived] Amass L, Li H, Gundapaneni BK, Schwartz JH, Keohane DJ. Influence of baseline neurologic severity on disease progression and the associated disease-modifying effects of tafamidis in patients with transthyretin amyloid polyneuropathy. Orphanet J Rare Dis. 2018 Dec 17;13(1):225. doi: 10.1186/s13023-018-0947-7. PMID 30558645
- [Derived] Barroso FA, Judge DP, Ebede B, Li H, Stewart M, Amass L, Sultan MB. Long-term safety and efficacy of tafamidis for the treatment of hereditary transthyretin amyloid polyneuropathy: results up to 6 years. Amyloid. 2017 Sep;24(3):194-204. doi: 10.1080/13506129.2017.1357545. Epub 2017 Jul 31. PMID 28758793
- [Derived] Waddington Cruz M, Amass L, Keohane D, Schwartz J, Li H, Gundapaneni B. Early intervention with tafamidis provides long-term (5.5-year) delay of neurologic progression in transthyretin hereditary amyloid polyneuropathy. Amyloid. 2016 Sep;23(3):178-183. doi: 10.1080/13506129.2016.1207163. Epub 2016 Aug 5. PMID 27494299
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=FX1A-303&StudyName=Safety%20And%20Efficacy%20Evaluation%20Of%20Fx-1006A%20In%20Subjects%20With%20Transthyretin%20Amyloidosis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled in B3461023 had transthyretin amyloid polyneuropathy (ATTR-PN), had not undergone liver/heart transplantation, and completed either B3461021 (Fx-006 [NCT00791492]: extension to Fx-005 [NCT00409175]) or B3461022 (Fx1A-201 [NCT00630864]). Val30Met (V30M): valine replaced by methionine in position 30 of TTR protein; NonVal30Met (NonV30M): TTR mutations other than V30M.
Pre-assignment Details: Prior to B3461023, V30M participants completed 18 months (M) blinded treatment (placebo or tafamidis) in Fx-005 followed by 12M tafamidis in Fx-006; nonV30M participants completed 12M tafamidis in Fx1A-201. Baseline (except treatment-emergent adverse events) was last measurement prior to 1st dose in Fx-005 (V30M) or Fx1A-201 (NonV30M). V30M:data from Baseline to M18 from Fx-005; after M18 to M30 from Fx-006; after M30 from B3461023. NonV30M:Baseline to M12 from Fx1A-201, after M12 from B3461023.
Groups:
- Val30Met: Tafamidis Then Tafamidis: Val30Met participants who received tafamidis in study B3461020 (Fx-005), continued the same in study B3461021 (Fx-006), received tafamidis 20 milligrams (mg) soft gelatin capsule orally once daily for up to 10 years from the date of enrollment in this study B3461023 (Fx1A-303) or until they had an access to tafamidis for ATTR-PN via prescription, upon regulatory approval in respective countries.
- Val30Met: Placebo Then Tafamidis: Val30Met participants who received placebo in study B3461020 (Fx-005) and assigned to receive tafamidis in study B3461021 (Fx-006) and study B3461023 (Fx1A-303), received tafamidis 20 mg soft gelatin capsule orally once daily for up to 10 years from the date of enrollment in this study B3461023 (Fx1A-303) or until they had an access to tafamidis for ATTR-PN via prescription, upon regulatory approval in respective countries.
- NonVal30Met: Tafamidis: NonVal30Met participants who received tafamidis in study B3461022 (Fx1A-201), received tafamidis 20 mg soft gelatin capsule orally once daily for up to 10 years from the date of enrollment in this study B3461023 (Fx1A-303) or until they had an access to tafamidis for ATTR-PN via prescription, upon regulatory approval in respective countries.
Period: Overall Study
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis
Started | 38 | 37 | 18
Treated | 38 | 37 | 18
Completed | 32 | 28 | 8
Not Completed | 6 | 9 | 10
Not completed — Other | 1 | 4 | 0
Not completed — Death | 1 | 1 | 5
Not completed — Adverse Event | 3 | 1 | 2
Not completed — Participant withdrew consent | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis | Total
Number analyzed (Participants) | 38 | 37 | 18 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 34 | 9 | 76
  >=65 years | 5 | 3 | 9 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 6 | 47
  Male | 18 | 16 | 12 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 33 | 34 | 17 | 84
  Latino American | 5 | 3 | 0 | 8
  Afro-Caribbean | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Val30Met Group: Neuropathy Impairment Score Lower Limb (NIS-LL) Score at Baseline
Description: NIS-LL: a subscale (of 37-item NIS questionnaire) that provided a total neuropathic deficit score for the lower limbs. It assess muscle weakness, reflexes, sensation; scored separately for left, right limbs. Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae); sensation (touch pressure, pin-prick, vibration, joint position) scored 0=normal, 1=decreased, or 2=absent. Total possible NIS-LL score range 0-88, high score=more impairment.
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461020 (Fx-005)
Population: ITT population included all enrolled participants who had taken at least one dose of study medication, and who had baseline and at least one post-baseline NIS-LL measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
units on a scale | 6.8 (10.8) | 11.6 (14.1)

2. Primary Outcome: Val30Met Group: Change From B3461020 Baseline in Neuropathy Impairment Score Lower Limb (NIS-LL) Score at Month 30
Description: as for outcome 1
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461020 (Fx-005), Month 30
Population: ITT population included all enrolled participants who had taken at least one dose of study medication, and who had baseline and at least one post-baseline NIS-LL measure. Here, "Overall number of participants analyzed " signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 36
units on a scale | 3.8 (1.5) | 6.4 (1.6)

3. Primary Outcome: Val30Met Group: Change From B3461020 Baseline in Neuropathy Impairment Score Lower Limb (NIS-LL) Score at Month 66
Description: as for outcome 1
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461020 (Fx-005), Month 66
Population: ITT population included all enrolled participants who had taken at least one dose of study medication, and who had baseline and at least one post-baseline NIS-LL measure. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 34 | 31
units on a scale | 7.8 (1.6) | 11.3 (1.6)

4. Primary Outcome: NonVal30Met Group: Neuropathy Impairment Score Lower Limb (NIS-LL) Score at Baseline
Description: as for outcome 1
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461022 (Fx1A-201)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale | 31.1 (24.4)

5. Primary Outcome: NonVal30Met Group: Change From B3461022 Baseline in Neuropathy Impairment Score Lower Limb (NIS-LL) Score at Month 12
Description: as for outcome 1
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461022 (Fx1A-201), Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale | 2.5 (2.0)

6. Primary Outcome: NonVal30Met Group: Change From B3461022 Baseline in Neuropathy Impairment Score Lower Limb (NIS-LL) Score at Month 60
Description: as for outcome 1
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461022 (Fx1A-201), Month 60
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 7
units on a scale | 12.0 (2.7)

7. Primary Outcome: Val30Met Group: Total Quality of Life (TQOL) Score Assessed Using Norfolk Quality of Life for Diabetic Neuropathy (QOL-DN) Questionnaire at Baseline
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire; assessed impact of DN on health related QOL of participants with DN. Scoring was based on 35 questions that yield a TQOL as well as 5 subscale scores: symptoms, activities of daily living (ADLs), large fiber neuropathy/physical functioning, small fiber neuropathy, and autonomic neuropathy. TQOL score: sum of all items, total possible score range= -2 to 138, where higher score=worse QOL.
Time Frame: Baseline of B3461020 (Fx-005)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 36
units on a scale | 24.1 (26.3) | 29.9 (30.1)

8. Primary Outcome: Val30Met Group: Change From B3461020 Baseline in Total Quality of Life (TQOL) Score Assessed Using Norfolk Quality of Life for Diabetic Neuropathy (QOL-DN) Questionnaire at Month 30
Description: as for outcome 7
Time Frame: Baseline of B3461020 (Fx-005), Month 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 37 | 36
units on a scale | 0.1 (3.3) | 4.5 (3.4)

9. Primary Outcome: Val30Met Group: Change From B3461020 Baseline in Total Quality of Life (TQOL) Score Assessed Using Norfolk Quality of Life for Diabetic Neuropathy (QOL-DN) Questionnaire at Month 66
Description: as for outcome 7
Time Frame: Baseline of B3461020 (Fx-005), Month 66
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 33 | 31
units on a scale | 5.2 (3.4) | 5.3 (3.5)

10. Primary Outcome: NonVal30Met Group: Total Quality of Life (TQOL) Score Assessed Using Norfolk Quality of Life for Diabetic Neuropathy (QOL-DN) Questionnaire at Baseline
Description: as for outcome 7
Time Frame: Baseline of B3461022 (Fx1A-201)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale | 53.9 (34.2)

11. Primary Outcome: NonVal30Met Group: Change From B3461022 Baseline in Total Quality of Life (TQOL) Score Assessed Using Norfolk Quality of Life for Diabetic Neuropathy (QOL-DN) Questionnaire at Month 12
Description: as for outcome 7
Time Frame: Baseline of B3461022 (Fx1A-201), Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale | 0.9 (5.7)

12. Primary Outcome: NonVal30Met Group: Change From B3461022 Baseline in Total Quality of Life (TQOL) Score Assessed Using Norfolk Quality of Life for Diabetic Neuropathy (QOL-DN) Questionnaire at Month 60
Description: as for outcome 7
Time Frame: Baseline of B3461022 (Fx1A-201), Month 60
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 7
units on a scale | 12.9 (7.4)

13. Primary Outcome: Val30Met Group: Karnofsky Performance Scale (KPS) Score at Month 30
Description: KPS: used for rating participant activities of daily living on 11-step scale from 0-100, higher score=participant is better able to carry out daily activities. Score range: 100=normal no complaints; no disease evidence, 90=able to carry normal activity; minor signs/symptoms of disease, 80=normal activity with effort; some signs/symptoms, 70=cares for self; unable to carry on normal activity, 60=requires occasional assistance, but able to care for most personal needs, 50=requires considerable assistance and frequent medical care, 40=disabled; requires special care, assistance, 30=severely disabled; hospital admission is indicated although death not imminent, 20=very sick; hospital admission necessary, 10=moribund; fatal processes progressing rapidly and 0=dead. The lower the score the worse is survival for most serious illnesses. Data for KPS score was not collected in parent studies Fx-005 and Fx-006, therefore not reported for any time points from parent studies.
Time Frame: Month 30 (Baseline of B3461023)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 37 | 36
units on a scale | 83.8 (12.99) | 80.3 (11.83)

14. Primary Outcome: Val30Met Group: Karnofsky Performance Scale (KPS) Score at Month 66
Description: as for outcome 13
Time Frame: Month 66 (Month 36 of B3461023)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 34 | 31
units on a scale | 85.9 (10.76) | 78.7 (17.65)

15. Primary Outcome: NonVal30Met Group: Karnofsky Performance Scale (KPS) Score at Baseline
Description: Karnofsky performance scale was used for rating participant activities of daily living. It rated participant on 11-step scale ranged from 0-100, higher score=participant is better able to carry out daily activities. The lower the score, the worse the survival for most serious illnesses. Score range: 100=normal no complaints; no evidence of disease, 90=able to carry on normal activity; minor signs/symptoms of disease, 80=normal activity with effort; some signs or symptoms, 70=cares for self; unable to carry on normal activity or to do active work, 60=requires occasional assistance, but able to care for most personal needs, 50=requires considerable assistance and frequent medical care, 40=disabled; requires special care and assistance, 30=severely disabled; hospital admission is indicated although death not imminent, 20=very sick; hospital admission necessary, 10=moribund; fatal processes progressing rapidly and 0=dead, where lower score=worse survival for most serious illnesses.
Time Frame: Baseline of B3461022 (Fx1A-201)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale | 72.2 (13.53)

16. Primary Outcome: NonVal30Met Group: Change From B3461022 Baseline in Karnofsky Performance Scale (KPS) Score at Month 12
Description: as for outcome 15
Time Frame: Baseline of B3461022 (Fx1A-201), Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale | -3.1 (2.57)

17. Primary Outcome: NonVal30Met Group: Change From B3461022 Baseline in Karnofsky Performance Scale (KPS) Score at Month 60
Description: as for outcome 15
Time Frame: Baseline of B3461022 (Fx1A-201), Month 60
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 7
units on a scale | -12.4 (3.73)

18. Primary Outcome: Val30Met Group: Number of Participants by Ambulation Stage at Baseline
Description: Ambulatory status for each Val30Met participant was collected using ambulatory data collection forms in [B3461020 (Fx-005), B3461021 (Fx-006)] or forms based on modified polyneuropathy disability (mPND) score in B3461023 (after protocol amendment 1.1). The data were categorized to 3 ambulation stages: Stage 1 (normal), Stage 2 (some assistance required), or Stage 3 (not ambulatory).
Time Frame: Baseline of B3461020 (Fx-005)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 37 | 36
Participants
  Stage 1 (Normal) | 37 | 36
  Stage 2 (Some assistance required) | 0 | 0
  Stage 3 (Not ambulatory) | 0 | 0

19. Primary Outcome: Val30Met Group: Number of Participants by Ambulation Stage at Month 30
Description: Ambulatory status for each Val30Met participant was collected using ambulatory data collection forms in [B3461020 (Fx-005), B3461021 (Fx-006)] or forms based on mPND score in B3461023 (after protocol amendment 1.1). The data were categorized to 3 ambulation stages: Stage 1 (normal), Stage 2 (some assistance required), or Stage 3 (not ambulatory).
Time Frame: Month 30
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 36
Participants
  Stage 1 (Normal) | 37 | 34
  Stage 2 (Some assistance required) | 0 | 1
  Stage 3 (Not ambulatory) | 1 | 1

20. Primary Outcome: Val30Met Group: Number of Participants by Ambulation Stage at Month 66
Description: as for outcome 19
Time Frame: Month 66
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 24 | 18
Participants
  Stage 1 (Normal) | 22 | 15
  Stage 2 (Some assistance required) | 2 | 3
  Stage 3 (Not ambulatory) | 0 | 0

21. Primary Outcome: NonVal30Met Group: Number of Participants by Ambulation Stage at Baseline
Description: Ambulatory status for each NonVal30Met participant was collected using ambulatory data collection forms in B3461022 (Fx1A-201) or forms based on mPND score in B3461023 (after protocol amendment 1.1). The data were categorized to 3 ambulation stages: Stage 1 (normal), Stage 2 (some assistance required), or Stage 3 (not ambulatory).
Time Frame: Baseline of B3461022 (Fx1A-201)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 12
Participants
  Stage 1 (Normal) | 7
  Stage 2 (Some assistance required) | 5
  Stage 3 (Not ambulatory) | 0

22. Primary Outcome: NonVal30Met Group: Number of Participants by Ambulation Stage at Month 12
Description: as for outcome 21
Time Frame: Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 13
Participants
  Stage 1 (Normal) | 7
  Stage 2 (Some assistance required) | 5
  Stage 3 (Not ambulatory) | 1

23. Primary Outcome: NonVal30Met Group: Number of Participants by Ambulation Stage at Month 60
Description: as for outcome 21
Time Frame: Month 60
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 7
Participants
  Stage 1 (Normal) | 1
  Stage 2 (Some assistance required) | 6
  Stage 3 (Not ambulatory) | 0

24. Secondary Outcome: Val30Met Group: Change From B3461020 Baseline in NIS-LL Score at Month 6, 12, 18, 24, 42, 54, 78, 90, 102, 114 and 126
Description: as for outcome 1
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461020 (Fx-005), Month 6, 12, 18, 24, 42, 54, 78, 90, 102, 114 and 126
Population: ITT population included all enrolled participants who had taken at least one dose of study medication, and who had baseline and at least one post-baseline NIS-LL measure. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
units on a scale
  NIS-LL: Change at Month 6 | 1.4 (1.5) | 0.6 (1.5)
  NIS-LL: Change at Month 12 | 1.4 (1.5) | 3.6 (1.5)
  NIS-LL: Change at Month 18 | 2.6 (1.5) | 4.4 (1.5)
  NIS-LL: Change at Month 24 | 3.4 (1.5) | 6.1 (1.5)
  NIS-LL: Change at Month 42: number analyzed (Participants) | 37 | 35
  NIS-LL: Change at Month 42 | 4.5 (1.5) | 8.9 (1.6)
  NIS-LL: Change at Month 54: number analyzed (Participants) | 36 | 34
  NIS-LL: Change at Month 54 | 6.3 (1.5) | 8.6 (1.6)
  NIS-LL: Change at Month 78: number analyzed (Participants) | 9 | 7
  NIS-LL: Change at Month 78 | 14.8 (2.4) | 9.8 (2.6)
  NIS-LL: Change at Month 90: number analyzed (Participants) | 9 | 6
  NIS-LL: Change at Month 90 | 17.1 (2.4) | 8.6 (2.8)
  NIS-LL: Change at Month 102: number analyzed (Participants) | 6 | 5
  NIS-LL: Change at Month 102 | 26.0 (2.8) | 12.5 (3.0)
  NIS-LL: Change at Month 114: number analyzed (Participants) | 4 | 4
  NIS-LL: Change at Month 114 | 22.0 (3.3) | 14.2 (3.3)
  NIS-LL: Change at Month 126: number analyzed (Participants) | 2 | 2
  NIS-LL: Change at Month 126 | 36.4 (4.6) | 12.6 (4.6)

25. Secondary Outcome: Val30Met Group: NIS-LL Subscales Scores: Muscle Weakness (MW), MW-Hip, MW-Knee, MW-Ankle, MW-Toe, NIS-LL Reflexes, NIS-LL Sensory at Baseline
Description: NIS-LL: a subscale (of 37-item NIS questionnaire) that provided a total neuropathic deficit score for the lower limbs. It assess muscle weakness, reflexes, sensation; scored separately for left, right limbs with a total possible NIS-LL score range of 0 to 88, higher score=greater impairment. Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae); sensation (touch pressure, pin-prick, vibration, joint position) scored 0=normal, 1=decreased, or 2=absent. NIS-LL Muscle Weakness score range is 0 to 64, high score=more impairment. NIS-LL Sensation score range is 0 to 16, high score=more impairment. NIS-LL Reflexes score range is 0 to 8, high score=more impairment.
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461020 (Fx-005)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
units on a scale
  NIS-LL MW: Baseline | 2.1 (6.4) | 4.2 (9.6)
  NIS-LL MW-Hip: Baseline | 0.2 (0.8) | 0.3 (1.1)
  NIS-LL MW-Knee: Baseline | 0.2 (0.9) | 0.4 (1.5)
  NIS-LL MW-Ankle: Baseline | 0.4 (1.5) | 1.3 (3.7)
  NIS-LL MW-Toe: Baseline | 1.3 (3.6) | 2.2 (4.2)
  NIS-LL Reflexes: Baseline | 0.8 (1.8) | 1.8 (2.4)
  NIS-LL Sensory: Baseline | 3.9 (3.7) | 5.6 (3.8)

26. Secondary Outcome: Val30Met Group: Change From B3461020 Baseline in NIS-LL Subscales Scores: Muscle Weakness (MW), MW-Hip, MW-Knee, MW-Ankle, MW-Toe, NIS-LL Reflexes, NIS-LL Sensory at Month 6, 12, 18, 24, 30, 42, 54, 66, 78, 90, 102, 114 and 126
Description: as for outcome 25
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461020 (Fx-005), Month 6, 12, 18, 24, 30, 42, 54, 66, 78, 90, 102, 114 and 126
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
units on a scale
  NIS-LL MW: Change at Month 6 | 0.6 (1.2) | 0.5 (1.2)
  NIS-LL MW: Change at Month 12 | 0.8 (1.2) | 2.4 (1.2)
  NIS-LL MW: Change at Month 18 | 1.3 (1.2) | 3.1 (1.2)
  NIS-LL MW: Change at Month 24 | 1.5 (1.2) | 4.0 (1.2)
  NIS-LL MW: Change at Month 30: number analyzed (Participants) | 38 | 36
  NIS-LL MW: Change at Month 30 | 2.5 (1.2) | 4.4 (1.2)
  NIS-LL MW: Change at Month 42: number analyzed (Participants) | 37 | 35
  NIS-LL MW: Change at Month 42 | 2.1 (1.2) | 6.3 (1.2)
  NIS-LL MW: Change at Month 54: number analyzed (Participants) | 36 | 34
  NIS-LL MW: Change at Month 54 | 3.1 (1.2) | 5.7 (1.2)
  NIS-LL MW: Change at Month 66: number analyzed (Participants) | 34 | 31
  NIS-LL MW: Change at Month 66 | 4.2 (1.2) | 7.4 (1.2)
  NIS-LL MW: Change at Month 78: number analyzed (Participants) | 9 | 7
  NIS-LL MW: Change at Month 78 | 8.7 (1.9) | 6.9 (2.1)
  NIS-LL MW: Change at Month 90: number analyzed (Participants) | 9 | 6
  NIS-LL MW: Change at Month 90 | 11.0 (1.9) | 5.4 (2.2)
  NIS-LL MW: Change at Month 102: number analyzed (Participants) | 6 | 5
  NIS-LL MW: Change at Month 102 | 18.2 (2.2) | 7.5 (2.4)
  NIS-LL MW: Change at Month 114: number analyzed (Participants) | 4 | 4
  NIS-LL MW: Change at Month 114 | 13.1 (2.6) | 9.1 (2.6)
  NIS-LL MW: Change at Month 126: number analyzed (Participants) | 2 | 2
  NIS-LL MW: Change at Month 126 | 27.9 (3.6) | 10.0 (3.6)
  NIS-LL MW-Hip: Change at Month 6 | 0.2 (0.3) | -0.1 (0.3)
  NIS-LL MW-Hip: Change at Month 12 | 0.2 (0.3) | 0.3 (0.3)
  NIS-LL MW-Hip: Change at Month 18 | 0.3 (0.3) | 0.3 (0.3)
  NIS-LL MW-Hip: Change at Month 24 | 0.4 (0.3) | 0.4 (0.3)
  NIS-LL MW-Hip: Change at Month 30: number analyzed (Participants) | 38 | 36
  NIS-LL MW-Hip: Change at Month 30 | 0.7 (0.3) | 0.7 (0.3)
  NIS-LL MW-Hip: Change at Month 42: number analyzed (Participants) | 37 | 35
  NIS-LL MW-Hip: Change at Month 42 | 0.4 (0.3) | 0.7 (0.3)
  NIS-LL MW-Hip: Change at Month 54: number analyzed (Participants) | 36 | 34
  NIS-LL MW-Hip: Change at Month 54 | 0.5 (0.3) | 0.4 (0.3)
  NIS-LL MW-Hip: Change at Month 66: number analyzed (Participants) | 34 | 31
  NIS-LL MW-Hip: Change at Month 66 | 0.5 (0.3) | 0.5 (0.3)
  NIS-LL MW-Hip: Change at Month 78: number analyzed (Participants) | 9 | 7
  NIS-LL MW-Hip: Change at Month 78 | 0.7 (0.5) | 0.1 (0.5)
  NIS-LL MW-Hip: Change at Month 90: number analyzed (Participants) | 9 | 6
  NIS-LL MW-Hip: Change at Month 90 | 0.9 (0.5) | 0.0 (0.6)
  NIS-LL MW-Hip: Change at Month 102: number analyzed (Participants) | 6 | 5
  NIS-LL MW-Hip: Change at Month 102 | 2.1 (0.6) | 0.0 (0.6)
  NIS-LL MW-Hip: Change at Month 114: number analyzed (Participants) | 4 | 4
  NIS-LL MW-Hip: Change at Month 114 | 0.4 (0.7) | 0.9 (0.7)
  NIS-LL MW-Hip: Change at Month 126: number analyzed (Participants) | 2 | 2
  NIS-LL MW-Hip: Change at Month 126 | 2.3 (0.9) | 2.2 (0.9)
  NIS-LL MW-Knee: Change at Month 6 | 0.1 (0.3) | 0.1 (0.3)
  NIS-LL MW-Knee: Change at Month 12 | 0.1 (0.3) | 0.4 (0.3)
  NIS-LL MW-Knee: Change at Month 18 | 0.2 (0.3) | 0.6 (0.3)
  NIS-LL MW-Knee: Change at Month 24 | 0.3 (0.3) | 0.4 (0.3)
  NIS-LL MW-Knee: Change at Month 30: number analyzed (Participants) | 38 | 36
  NIS-LL MW-Knee: Change at Month 30 | 0.6 (0.3) | 0.6 (0.3)
  NIS-LL MW-Knee: Change at Month 42: number analyzed (Participants) | 37 | 35
  NIS-LL MW-Knee: Change at Month 42 | 0.4 (0.3) | 0.7 (0.3)
  NIS-LL MW-Knee: Change at Month 54: number analyzed (Participants) | 36 | 34
  NIS-LL MW-Knee: Change at Month 54 | 0.5 (0.3) | 0.4 (0.3)
  NIS-LL MW-Knee: Change at Month 66: number analyzed (Participants) | 34 | 31
  NIS-LL MW-Knee: Change at Month 66 | 0.4 (0.3) | 0.7 (0.3)
  NIS-LL MW-Knee: Change at Month 78: number analyzed (Participants) | 9 | 7
  NIS-LL MW-Knee: Change at Month 78 | 0.5 (0.5) | 1.0 (0.5)
  NIS-LL MW-Knee: Change at Month 90: number analyzed (Participants) | 9 | 6
  NIS-LL MW-Knee: Change at Month 90 | 1.6 (0.5) | 0.5 (0.6)
  NIS-LL MW-Knee: Change at Month 102: number analyzed (Participants) | 6 | 5
  NIS-LL MW-Knee: Change at Month 102 | 5.1 (0.5) | 1.1 (0.6)
  NIS-LL MW-Knee: Change at Month 114: number analyzed (Participants) | 4 | 4
  NIS-LL MW-Knee: Change at Month 114 | 0.4 (0.7) | 1.4 (0.7)
  NIS-LL MW-Knee: Change at Month 126: number analyzed (Participants) | 2 | 2
  NIS-LL MW-Knee: Change at Month 126 | 3.2 (0.9) | 3.7 (0.9)
  NIS-LL MW-Ankle: Change at Month 6 | 0.2 (0.5) | 0.3 (0.5)
  NIS-LL MW-Ankle: Change at Month 12 | 0.4 (0.5) | 0.7 (0.5)
  NIS-LL MW-Ankle: Change at Month 18 | 0.5 (0.5) | 1.1 (0.5)
  NIS-LL MW-Ankle: Change at Month 24 | 0.5 (0.5) | 1.6 (0.5)
  NIS-LL MW-Ankle: Change at Month 30: number analyzed (Participants) | 38 | 36
  NIS-LL MW-Ankle: Change at Month 30 | 0.8 (0.5) | 1.4 (0.5)
  NIS-LL MW-Ankle: Change at Month 42: number analyzed (Participants) | 37 | 35
  NIS-LL MW-Ankle: Change at Month 42 | 0.8 (0.5) | 2.3 (0.5)
  NIS-LL MW-Ankle: Change at Month 54: number analyzed (Participants) | 36 | 34
  NIS-LL MW-Ankle: Change at Month 54 | 1.2 (0.5) | 2.0 (0.5)
  NIS-LL MW-Ankle: Change at Month 66: number analyzed (Participants) | 34 | 31
  NIS-LL MW-Ankle: Change at Month 66 | 1.6 (0.5) | 2.8 (0.5)
  NIS-LL MW-Ankle: Change at Month 78: number analyzed (Participants) | 9 | 7
  NIS-LL MW-Ankle: Change at Month 78 | 3.5 (0.7) | 2.5 (0.8)
  NIS-LL MW-Ankle: Change at Month 90: number analyzed (Participants) | 9 | 6
  NIS-LL MW-Ankle: Change at Month 90 | 3.9 (0.7) | 2.6 (0.9)
  NIS-LL MW-Ankle: Change at Month 102: number analyzed (Participants) | 6 | 5
  NIS-LL MW-Ankle: Change at Month 102 | 5.8 (0.9) | 3.2 (1.0)
  NIS-LL MW-Ankle: Change at Month 114: number analyzed (Participants) | 4 | 4
  NIS-LL MW-Ankle: Change at Month 114 | 5.1 (1.0) | 3.7 (1.1)
  NIS-LL MW-Ankle: Change at Month 126: number analyzed (Participants) | 2 | 2
  NIS-LL MW-Ankle: Change at Month 126 | 10.8 (1.4) | 2.1 (1.4)
  NIS-LL MW-Toe: Change at Month 6 | -0.1 (0.5) | 0.3 (0.5)
  NIS-LL MW-Toe: Change at Month 12 | -0.1 (0.5) | 1.2 (0.5)
  NIS-LL MW-Toe: Change at Month 18 | 0.2 (0.5) | 1.3 (0.5)
  NIS-LL MW-Toe: Change at Month 24 | 0.1 (0.5) | 1.8 (0.5)
  NIS-LL MW-Toe: Change at Month 30: number analyzed (Participants) | 38 | 36
  NIS-LL MW-Toe: Change at Month 30 | 0.3 (0.5) | 1.9 (0.5)
  NIS-LL MW-Toe: Change at Month 42: number analyzed (Participants) | 37 | 35
  NIS-LL MW-Toe: Change at Month 42 | 0.3 (0.5) | 2.7 (0.5)
  NIS-LL MW-Toe: Change at Month 54: number analyzed (Participants) | 36 | 34
  NIS-LL MW-Toe: Change at Month 54 | 0.6 (0.5) | 2.9 (0.5)
  NIS-LL MW-Toe: Change at Month 66: number analyzed (Participants) | 34 | 31
  NIS-LL MW-Toe: Change at Month 66 | 1.5 (0.5) | 3.6 (0.5)
  NIS-LL MW-Toe: Change at Month 78: number analyzed (Participants) | 9 | 7
  NIS-LL MW-Toe: Change at Month 78 | 3.9 (0.8) | 3.5 (0.9)
  NIS-LL MW-Toe: Change at Month 90: number analyzed (Participants) | 9 | 6
  NIS-LL MW-Toe: Change at Month 90 | 4.5 (0.8) | 2.5 (1.0)
  NIS-LL MW-Toe: Change at Month 102: number analyzed (Participants) | 6 | 5
  NIS-LL MW-Toe: Change at Month 102 | 5.1 (0.9) | 3.4 (1.0)
  NIS-LL MW-Toe: Change at Month 114: number analyzed (Participants) | 4 | 4
  NIS-LL MW-Toe: Change at Month 114 | 7.0 (1.1) | 3.3 (1.1)
  NIS-LL MW-Toe: Change at Month 126: number analyzed (Participants) | 2 | 2
  NIS-LL MW-Toe: Change at Month 126 | 11.4 (1.5) | 2.4 (1.5)
  NIS-LL Reflexes: Change at Month 6 | 0.2 (0.2) | 0.1 (0.2)
  NIS-LL Reflexes: Change at Month 12 | 0.4 (0.2) | 0.5 (0.2)
  NIS-LL Reflexes: Change at Month 18 | 0.4 (0.2) | 0.5 (0.2)
  NIS-LL Reflexes: Change at Month 24 | 0.7 (0.2) | 0.9 (0.2)
  NIS-LL Reflexes: Change at Month 30: number analyzed (Participants) | 38 | 36
  NIS-LL Reflexes: Change at Month 30 | 0.5 (0.2) | 0.7 (0.2)
  NIS-LL Reflexes: Change at Month 42: number analyzed (Participants) | 37 | 35
  NIS-LL Reflexes: Change at Month 42 | 0.7 (0.2) | 1.0 (0.2)
  NIS-LL Reflexes: Change at Month 54: number analyzed (Participants) | 36 | 34
  NIS-LL Reflexes: Change at Month 54 | 0.9 (0.2) | 1.2 (0.2)
  NIS-LL Reflexes: Change at Month 66: number analyzed (Participants) | 34 | 31
  NIS-LL Reflexes: Change at Month 66 | 1.1 (0.2) | 1.4 (0.2)
  NIS-LL Reflexes: Change at Month 78: number analyzed (Participants) | 9 | 7
  NIS-LL Reflexes: Change at Month 78 | 1.5 (0.4) | 1.3 (0.4)
  NIS-LL Reflexes: Change at Month 90: number analyzed (Participants) | 9 | 6
  NIS-LL Reflexes: Change at Month 90 | 1.4 (0.4) | 0.7 (0.5)
  NIS-LL Reflexes: Change at Month 102: number analyzed (Participants) | 6 | 5
  NIS-LL Reflexes: Change at Month 102 | 2.0 (0.5) | 1.5 (0.5)
  NIS-LL Reflexes: Change at Month 114: number analyzed (Participants) | 4 | 4
  NIS-LL Reflexes: Change at Month 114 | 3.0 (0.6) | 2.9 (0.6)
  NIS-LL Reflexes: Change at Month 126: number analyzed (Participants) | 2 | 2
  NIS-LL Reflexes: Change at Month 126 | 3.6 (0.8) | 1.1 (0.8)
  NIS-LL Sensory: Change at Month 6 | 0.4 (0.5) | 0.4 (0.5)
  NIS-LL Sensory: Change at Month 12 | -0.1 (0.5) | 1.1 (0.5)
  NIS-LL Sensory: Change at Month 18 | 0.6 (0.5) | 1.3 (0.5)
  NIS-LL Sensory: Change at Month 24 | 0.9 (0.5) | 1.6 (0.5)
  NIS-LL Sensory: Change at Month 30: number analyzed (Participants) | 38 | 36
  NIS-LL Sensory: Change at Month 30 | 0.5 (0.5) | 1.7 (0.5)
  NIS-LL Sensory: Change at Month 42: number analyzed (Participants) | 37 | 35
  NIS-LL Sensory: Change at Month 42 | 1.4 (0.5) | 2.0 (0.5)
  NIS-LL Sensory: Change at Month 54: number analyzed (Participants) | 36 | 34
  NIS-LL Sensory: Change at Month 54 | 2.0 (0.5) | 2.1 (0.6)
  NIS-LL Sensory: Change at Month 66: number analyzed (Participants) | 34 | 31
  NIS-LL Sensory: Change at Month 66 | 2.2 (0.5) | 2.9 (0.6)
  NIS-LL Sensory: Change at Month 78: number analyzed (Participants) | 9 | 7
  NIS-LL Sensory: Change at Month 78 | 4.3 (0.8) | 1.9 (0.9)
  NIS-LL Sensory: Change at Month 90: number analyzed (Participants) | 9 | 6
  NIS-LL Sensory: Change at Month 90 | 4.5 (0.8) | 2.8 (0.9)
  NIS-LL Sensory: Change at Month 102: number analyzed (Participants) | 6 | 5
  NIS-LL Sensory: Change at Month 102 | 5.5 (0.9) | 3.9 (1.0)
  NIS-LL Sensory: Change at Month 114: number analyzed (Participants) | 4 | 4
  NIS-LL Sensory: Change at Month 114 | 5.4 (1.1) | 2.6 (1.1)
  NIS-LL Sensory: Change at Month 126: number analyzed (Participants) | 2 | 2
  NIS-LL Sensory: Change at Month 126 | 4.6 (1.5) | 1.8 (1.5)

27. Secondary Outcome: NonVal30Met Group: Change From B3461022 Baseline in NIS-LL Score at Month 6, 24, 36, 48, 72, 84, 96, 108 and 120
Description: as for outcome 1
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461022 (Fx1A-201), 6, 24, 36, 48, 72, 84, 96, 108 and 120
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale
  NIS-LL: Change at Month 6 | -0.7 (2.0)
  NIS-LL: Change at Month 24 | 6.6 (2.0)
  NIS-LL: Change at Month 36: number analyzed (Participants) | 11
  NIS-LL: Change at Month 36 | 10.9 (2.3)
  NIS-LL: Change at Month 48: number analyzed (Participants) | 10
  NIS-LL: Change at Month 48 | 12.3 (2.4)
  NIS-LL: Change at Month 72: number analyzed (Participants) | 3
  NIS-LL: Change at Month 72 | 14.6 (3.7)
  NIS-LL: Change at Month 84: number analyzed (Participants) | 2
  NIS-LL: Change at Month 84 | 10.4 (4.4)
  NIS-LL: Change at Month 96: number analyzed (Participants) | 2
  NIS-LL: Change at Month 96 | 13.9 (4.4)
  NIS-LL: Change at Month 108: number analyzed (Participants) | 2
  NIS-LL: Change at Month 108 | 12.9 (4.4)
  NIS-LL: Change at Month 120: number analyzed (Participants) | 2
  NIS-LL: Change at Month 120 | 13.9 (4.4)

28. Secondary Outcome: NonVal30Met Group: NIS-LL Subscales Scores: Muscle Weakness (MW), MW-Hip, MW-Knee, MW-Ankle, MW-Toe, NIS-LL Reflexes, NIS-LL Sensory at Baseline
Description: as for outcome 25
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461022 (Fx1A-201)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale
  NIS-LL MW: Baseline | 16.6 (16.9)
  NIS-LL MW-Hip: Baseline | 1.6 (2.4)
  NIS-LL MW-Knee: Baseline | 2.5 (3.8)
  NIS-LL MW-Ankle: Baseline | 5.5 (6.0)
  NIS-LL MW-Toe: Baseline | 6.9 (6.6)
  NIS-LL Reflexes: Baseline | 5.6 (3.4)
  NIS-LL Sensory: Baseline | 8.9 (5.4)

29. Secondary Outcome: NonVal30Met Group: Change From B3461022 Baseline in NIS-LL Subscales Scores: Muscle Weakness (MW), MW-Hip, MW-Knee, MW-Ankle, MW-Toe, NIS-LL Reflexes, NIS-LL Sensory at Month 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120
Description: as for outcome 25
Time Frame: Baseline (i.e. last measurement prior to first dose) of B3461022 (Fx1A-201), Month 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale
  NIS-LL MW: Change at Month 6 | -0.4 (1.5)
  NIS-LL MW: Change at Month 12 | 2.3 (1.5)
  NIS-LL MW: Change at Month 24 | 5.1 (1.5)
  NIS-LL MW: Change at Month 36: number analyzed (Participants) | 11
  NIS-LL MW: Change at Month 36 | 7.3 (1.8)
  NIS-LL MW: Change at Month 48: number analyzed (Participants) | 10
  NIS-LL MW: Change at Month 48 | 9.7 (1.9)
  NIS-LL MW: Change at Month 60: number analyzed (Participants) | 7
  NIS-LL MW: Change at Month 60 | 8.0 (2.1)
  NIS-LL MW: Change at Month 72: number analyzed (Participants) | 3
  NIS-LL MW: Change at Month 72 | 8.1 (3.0)
  NIS-LL MW: Change at Month 84: number analyzed (Participants) | 2
  NIS-LL MW: Change at Month 84 | 5.7 (3.6)
  NIS-LL MW: Change at Month 96: number analyzed (Participants) | 2
  NIS-LL MW: Change at Month 96 | 5.2 (3.6)
  NIS-LL MW: Change at Month 108: number analyzed (Participants) | 2
  NIS-LL MW: Change at Month 108 | 6.2 (3.6)
  NIS-LL MW: Change at Month 120: number analyzed (Participants) | 2
  NIS-LL MW: Change at Month 120 | 10.2 (3.6)
  NIS-LL MW-Hip: Change at Month 6 | -0.3 (0.6)
  NIS-LL MW-Hip: Change at Month 12 | 0.6 (0.6)
  NIS-LL MW-Hip: Change at Month 24 | 1.1 (0.6)
  NIS-LL MW-Hip: Change at Month 36: number analyzed (Participants) | 11
  NIS-LL MW-Hip: Change at Month 36 | 0.9 (0.6)
  NIS-LL MW-Hip: Change at Month 48: number analyzed (Participants) | 10
  NIS-LL MW-Hip: Change at Month 48 | 1.3 (0.6)
  NIS-LL MW-Hip: Change at Month 60: number analyzed (Participants) | 7
  NIS-LL MW-Hip: Change at Month 60 | 0.0 (0.7)
  NIS-LL MW-Hip: Change at Month 72: number analyzed (Participants) | 3
  NIS-LL MW-Hip: Change at Month 72 | 0.4 (0.9)
  NIS-LL MW-Hip: Change at Month 84: number analyzed (Participants) | 2
  NIS-LL MW-Hip: Change at Month 84 | 1.4 (1.0)
  NIS-LL MW-Hip: Change at Month 96: number analyzed (Participants) | 2
  NIS-LL MW-Hip: Change at Month 96 | 0.4 (1.0)
  NIS-LL MW-Hip: Change at Month 108: number analyzed (Participants) | 2
  NIS-LL MW-Hip: Change at Month 108 | 0.4 (1.0)
  NIS-LL MW-Hip: Change at Month 120: number analyzed (Participants) | 2
  NIS-LL MW-Hip: Change at Month 120 | 1.9 (1.0)
  NIS-LL MW-Knee: Change at Month 6 | 0.0 (0.7)
  NIS-LL MW-Knee: Change at Month 12 | 0.6 (0.7)
  NIS-LL MW-Knee: Change at Month 24 | 1.3 (0.7)
  NIS-LL MW-Knee: Change at Month 36: number analyzed (Participants) | 11
  NIS-LL MW-Knee: Change at Month 36 | 1.3 (0.8)
  NIS-LL MW-Knee: Change at Month 48: number analyzed (Participants) | 10
  NIS-LL MW-Knee: Change at Month 48 | 1.8 (0.8)
  NIS-LL MW-Knee: Change at Month 60: number analyzed (Participants) | 7
  NIS-LL MW-Knee: Change at Month 60 | -0.2 (0.9)
  NIS-LL MW-Knee: Change at Month 72: number analyzed (Participants) | 3
  NIS-LL MW-Knee: Change at Month 72 | 1.3 (1.1)
  NIS-LL MW-Knee: Change at Month 84: number analyzed (Participants) | 2
  NIS-LL MW-Knee: Change at Month 84 | 0.7 (1.3)
  NIS-LL MW-Knee: Change at Month 96: number analyzed (Participants) | 2
  NIS-LL MW-Knee: Change at Month 96 | 0.7 (1.3)
  NIS-LL MW-Knee: Change at Month 108: number analyzed (Participants) | 2
  NIS-LL MW-Knee: Change at Month 108 | 0.7 (1.3)
  NIS-LL MW-Knee: Change at Month 120: number analyzed (Participants) | 2
  NIS-LL MW-Knee: Change at Month 120 | 0.7 (1.3)
  NIS-LL MW-Ankle: Change at Month 6 | -0.2 (0.6)
  NIS-LL MW-Ankle: Change at Month 12 | 0.7 (0.6)
  NIS-LL MW-Ankle: Change at Month 24 | 1.5 (0.6)
  NIS-LL MW-Ankle: Change at Month 36: number analyzed (Participants) | 11
  NIS-LL MW-Ankle: Change at Month 36 | 2.7 (0.7)
  NIS-LL MW-Ankle: Change at Month 48: number analyzed (Participants) | 10
  NIS-LL MW-Ankle: Change at Month 48 | 3.3 (0.7)
  NIS-LL MW-Ankle: Change at Month 60: number analyzed (Participants) | 7
  NIS-LL MW-Ankle: Change at Month 60 | 4.6 (0.8)
  NIS-LL MW-Ankle: Change at Month 72: number analyzed (Participants) | 3
  NIS-LL MW-Ankle: Change at Month 72 | 2.8 (1.2)
  NIS-LL MW-Ankle: Change at Month 84: number analyzed (Participants) | 2
  NIS-LL MW-Ankle: Change at Month 84 | 2.0 (1.4)
  NIS-LL MW-Ankle: Change at Month 96: number analyzed (Participants) | 2
  NIS-LL MW-Ankle: Change at Month 96 | 2.0 (1.4)
  NIS-LL MW-Ankle: Change at Month 108: number analyzed (Participants) | 2
  NIS-LL MW-Ankle: Change at Month 108 | 2.0 (1.4)
  NIS-LL MW-Ankle: Change at Month 120: number analyzed (Participants) | 2
  NIS-LL MW-Ankle: Change at Month 120 | 2.0 (1.4)
  NIS-LL MW-Toe: Change at Month 6 | 0.5 (0.7)
  NIS-LL MW-Toe: Change at Month 12 | 0.8 (0.7)
  NIS-LL MW-Toe: Change at Month 24 | 1.5 (0.7)
  NIS-LL MW-Toe: Change at Month 36: number analyzed (Participants) | 11
  NIS-LL MW-Toe: Change at Month 36 | 2.6 (0.8)
  NIS-LL MW-Toe: Change at Month 48: number analyzed (Participants) | 10
  NIS-LL MW-Toe: Change at Month 48 | 3.5 (0.8)
  NIS-LL MW-Toe: Change at Month 60: number analyzed (Participants) | 7
  NIS-LL MW-Toe: Change at Month 60 | 3.9 (0.9)
  NIS-LL MW-Toe: Change at Month 72: number analyzed (Participants) | 3
  NIS-LL MW-Toe: Change at Month 72 | 3.8 (1.3)
  NIS-LL MW-Toe: Change at Month 84: number analyzed (Participants) | 2
  NIS-LL MW-Toe: Change at Month 84 | 1.7 (1.6)
  NIS-LL MW-Toe: Change at Month 96: number analyzed (Participants) | 2
  NIS-LL MW-Toe: Change at Month 96 | 2.2 (1.6)
  NIS-LL MW-Toe: Change at Month 108: number analyzed (Participants) | 2
  NIS-LL MW-Toe: Change at Month 108 | 3.2 (1.6)
  NIS-LL MW-Toe: Change at Month 120: number analyzed (Participants) | 2
  NIS-LL MW-Toe: Change at Month 120 | 5.7 (1.6)
  NIS-LL Reflexes: Change at Month 6 | -0.1 (0.4)
  NIS-LL Reflexes: Change at Month 12 | -0.2 (0.4)
  NIS-LL Reflexes: Change at Month 24 | 0.8 (0.4)
  NIS-LL Reflexes: Change at Month 36: number analyzed (Participants) | 11
  NIS-LL Reflexes: Change at Month 36 | 1.6 (0.5)
  NIS-LL Reflexes: Change at Month 48: number analyzed (Participants) | 10
  NIS-LL Reflexes: Change at Month 48 | 1.1 (0.5)
  NIS-LL Reflexes: Change at Month 60: number analyzed (Participants) | 7
  NIS-LL Reflexes: Change at Month 60 | 0.7 (0.6)
  NIS-LL Reflexes: Change at Month 72: number analyzed (Participants) | 3
  NIS-LL Reflexes: Change at Month 72 | 2.3 (0.9)
  NIS-LL Reflexes: Change at Month 84: number analyzed (Participants) | 2
  NIS-LL Reflexes: Change at Month 84 | 1.8 (1.1)
  NIS-LL Reflexes: Change at Month 96: number analyzed (Participants) | 2
  NIS-LL Reflexes: Change at Month 96 | 2.3 (1.1)
  NIS-LL Reflexes: Change at Month 108: number analyzed (Participants) | 2
  NIS-LL Reflexes: Change at Month 108 | 2.3 (1.1)
  NIS-LL Reflexes: Change at Month 120: number analyzed (Participants) | 2
  NIS-LL Reflexes: Change at Month 120 | -2.2 (1.1)
  NIS-LL Sensory: Change at Month 6 | -0.1 (0.7)
  NIS-LL Sensory: Change at Month 12 | 0.4 (0.7)
  NIS-LL Sensory: Change at Month 24 | 0.9 (0.7)
  NIS-LL Sensory: Change at Month 36: number analyzed (Participants) | 11
  NIS-LL Sensory: Change at Month 36 | 2.1 (0.8)
  NIS-LL Sensory: Change at Month 48: number analyzed (Participants) | 10
  NIS-LL Sensory: Change at Month 48 | 1.7 (0.8)
  NIS-LL Sensory: Change at Month 60: number analyzed (Participants) | 7
  NIS-LL Sensory: Change at Month 60 | 3.4 (0.9)
  NIS-LL Sensory: Change at Month 72: number analyzed (Participants) | 3
  NIS-LL Sensory: Change at Month 72 | 4.2 (1.2)
  NIS-LL Sensory: Change at Month 84: number analyzed (Participants) | 2
  NIS-LL Sensory: Change at Month 84 | 2.9 (1.4)
  NIS-LL Sensory: Change at Month 96: number analyzed (Participants) | 2
  NIS-LL Sensory: Change at Month 96 | 6.4 (1.4)
  NIS-LL Sensory: Change at Month 108: number analyzed (Participants) | 2
  NIS-LL Sensory: Change at Month 108 | 4.4 (1.4)
  NIS-LL Sensory: Change at Month 120: number analyzed (Participants) | 2
  NIS-LL Sensory: Change at Month 120 | 5.9 (1.4)

30. Secondary Outcome: Val30Met Group: Change From B3461020 Baseline in Total Quality of Life (TQOL) Score Assessed Using Norfolk Quality of Life for Diabetic Neuropathy (QOL-DN) Questionnaire at Month 6, 12, 18, 24, 42, 54, 78, 90, 102, 114, 126, 138
Description: as for outcome 7
Time Frame: Baseline of B3461020 (Fx-005), Month 6, 12, 18, 24, 42, 54, 78, 90, 102, 114, 126, 138
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
units on a scale
  TQOL: Change at Month 6: number analyzed (Participants) | 38 | 36
  TQOL: Change at Month 6 | -2.2 (3.3) | -0.5 (3.4)
  TQOL: Change at Month 12: number analyzed (Participants) | 38 | 36
  TQOL: Change at Month 12 | -2.8 (3.3) | 5.4 (3.4)
  TQOL: Change at Month 18: number analyzed (Participants) | 38 | 36
  TQOL: Change at Month 18 | -2.3 (3.3) | 6.4 (3.4)
  TQOL: Change at Month 24: number analyzed (Participants) | 38 | 36
  TQOL: Change at Month 24 | -3.2 (3.3) | 2.0 (3.4)
  TQOL: Change at Month 42: number analyzed (Participants) | 36 | 33
  TQOL: Change at Month 42 | 3.2 (3.3) | 1.8 (3.4)
  TQOL: Change at Month 54: number analyzed (Participants) | 36 | 33
  TQOL: Change at Month 54 | 3.0 (3.3) | 2.1 (3.4)
  TQOL: Change at Month 78: number analyzed (Participants) | 9 | 6
  TQOL: Change at Month 78 | 7.0 (4.8) | -3.9 (5.6)
  TQOL: Change at Month 90: number analyzed (Participants) | 7 | 5
  TQOL: Change at Month 90 | 3.2 (5.2) | -2.0 (6.0)
  TQOL: Change at Month 102: number analyzed (Participants) | 5 | 4
  TQOL: Change at Month 102 | 15.8 (5.9) | -7.3 (6.5)
  TQOL: Change at Month 114: number analyzed (Participants) | 4 | 4
  TQOL: Change at Month 114 | 18.9 (6.5) | -9.0 (6.5)
  TQOL: Change at Month 126: number analyzed (Participants) | 2 | 2
  TQOL: Change at Month 126 | 48.1 (8.7) | 2.0 (8.7)
  TQOL: Change at Month 138: number analyzed (Participants) | 1 | 1
  TQOL: Change at Month 138 | 55.4 (12.0) | 26.0 (12.0)

31. Secondary Outcome: Val30Met Group: TQOL Subscale Scores: Symptom, ADLs, Physical Functioning/Large Fiber Neuropathy, Small Fiber Neuropathy, Autonomic Neuropathy Assessed Using Norfolk QOL-DN at Baseline
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire to assess impact of DN on QOL; Item 1 to 7: scored as 1=symptom present, 0=symptom absent. Items 8 to 35: scored on 5-point Likert scale: 0=no problem to 4=severe problem (except item 32, where -1="somewhat better", -2=much better, 0=about the same, 1=somewhat worse, 2=much worse). Norfolk QOL-DN summarized in 5 domains (score range): physical functioning/large fiber neuropathy (-2 to 58), activities of daily living (ADLs) (0 to 20), symptoms (0 to 32), small fiber neuropathy (0 to 16), autonomic neuropathy (0 to 12); higher score=greater impairment, for each. Total score= -2 to 138 (higher score=worse QOL).
Time Frame: Baseline of B3461020 (Fx-005)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
units on a scale
  Symptom: Baseline: number analyzed (Participants) | 38 | 36
  Symptom: Baseline | 6.4 (5.4) | 6.8 (6.5)
  ADLs: Baseline: number analyzed (Participants) | 38 | 36
  ADLs: Baseline | 1.4 (3.5) | 1.9 (4.6)
  Physical Functioning/Large Fiber Neuropathy: Baseline: number analyzed (Participants) | 38 | 36
  Physical Functioning/Large Fiber Neuropathy: Baseline | 12.4 (14.4) | 15.9 (15.9)
  Small Fiber Neuropathy: Baseline: number analyzed (Participants) | 38 | 36
  Small Fiber Neuropathy: Baseline | 1.8 (3.2) | 3.1 (4.2)
  Autonomic Neuropathy: Baseline: number analyzed (Participants) | 38 | 36
  Autonomic Neuropathy: Baseline | 2.1 (2.8) | 2.2 (2.8)

32. Secondary Outcome: Val30Met:Change From Baseline in TQOL Subscale Scores:Symptom, ADLs, Physical Functioning/Large Fiber Neuropathy, Small Fiber Neuropathy, Autonomic Neuropathy Assessed Using Norfolk QOL-DN at Month 6, 12, 18, 24, 30, 42, 54, 66, 78, 90, 102, 114, 126, 138
Description: as for outcome 31
Time Frame: Baseline of B3461020 (Fx-005), Month 6, 12, 18, 24, 30, 42, 54, 66, 78, 90, 102, 114, 126 and 138
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
units on a scale
  Symptom: Change at Month 6: number analyzed (Participants) | 38 | 36
  Symptom: Change at Month 6 | -0.2 (0.8) | -0.1 (0.8)
  Symptom: Change at Month 12: number analyzed (Participants) | 38 | 36
  Symptom: Change at Month 12 | -0.9 (0.8) | 1.5 (0.8)
  Symptom: Change at Month 18: number analyzed (Participants) | 38 | 36
  Symptom: Change at Month 18 | -1.1 (0.8) | 0.6 (0.8)
  Symptom: Change at Month 24: number analyzed (Participants) | 37 | 36
  Symptom: Change at Month 24 | -1.1 (0.8) | 0.1 (0.8)
  Symptom: Change at Month 30: number analyzed (Participants) | 37 | 36
  Symptom: Change at Month 30 | -1.4 (0.8) | -0.7 (0.8)
  Symptom: Change at Month 42: number analyzed (Participants) | 36 | 33
  Symptom: Change at Month 42 | -0.4 (0.8) | -0.9 (0.8)
  Symptom: Change at Month 54: number analyzed (Participants) | 36 | 33
  Symptom: Change at Month 54 | -0.3 (0.8) | 0.2 (0.8)
  Symptom: Change at Month 66: number analyzed (Participants) | 33 | 31
  Symptom: Change at Month 66 | 0.6 (0.8) | -0.4 (0.8)
  Symptom: Change at Month 78: number analyzed (Participants) | 9 | 6
  Symptom: Change at Month 78 | 0.0 (1.2) | -2.8 (1.5)
  Symptom: Change at Month 90: number analyzed (Participants) | 7 | 5
  Symptom: Change at Month 90 | 1.0 (1.4) | -2.0 (1.6)
  Symptom: Change at Month 102: number analyzed (Participants) | 5 | 4
  Symptom: Change at Month 102 | -0.7 (1.6) | -2.8 (1.7)
  Symptom: Change at Month 114: number analyzed (Participants) | 4 | 4
  Symptom: Change at Month 114 | 1.9 (1.7) | -3.5 (1.7)
  Symptom: Change at Month 126: number analyzed (Participants) | 2 | 2
  Symptom: Change at Month 126 | 5.7 (2.4) | -1.3 (2.4)
  Symptom: Change at Month 138: number analyzed (Participants) | 1 | 1
  Symptom: Change at Month 138 | 4.1 (3.3) | 3.9 (3.3)
  ADLs: Change at Month 6: number analyzed (Participants) | 38 | 36
  ADLs: Change at Month 6 | 0.0 (0.6) | 0.2 (0.6)
  ADLs: Change at Month 12: number analyzed (Participants) | 38 | 36
  ADLs: Change at Month 12 | 0.7 (0.6) | 0.9 (0.6)
  ADLs: Change at Month 18: number analyzed (Participants) | 38 | 36
  ADLs: Change at Month 18 | 1.0 (0.6) | 1.3 (0.6)
  ADLs: Change at Month 24: number analyzed (Participants) | 38 | 36
  ADLs: Change at Month 24 | 0.7 (0.6) | 1.0 (0.6)
  ADLs: Change at Month 30: number analyzed (Participants) | 37 | 36
  ADLs: Change at Month 30 | 1.1 (0.6) | 1.2 (0.6)
  ADLs: Change at Month 42: number analyzed (Participants) | 36 | 33
  ADLs: Change at Month 42 | 1.5 (0.6) | 1.4 (0.6)
  ADLs: Change at Month 54: number analyzed (Participants) | 36 | 33
  ADLs: Change at Month 54 | 0.9 (0.6) | 1.1 (0.6)
  ADLs: Change at Month 66: number analyzed (Participants) | 33 | 31
  ADLs: Change at Month 66 | 1.5 (0.6) | 2.0 (0.6)
  ADLs: Change at Month 78: number analyzed (Participants) | 9 | 6
  ADLs: Change at Month 78 | 2.3 (0.9) | 1.2 (1.0)
  ADLs: Change at Month 90: number analyzed (Participants) | 7 | 5
  ADLs: Change at Month 90 | 1.7 (0.9) | 0.6 (1.1)
  ADLs: Change at Month 102: number analyzed (Participants) | 5 | 4
  ADLs: Change at Month 102 | 5.6 (1.1) | -0.8 (1.2)
  ADLs: Change at Month 114: number analyzed (Participants) | 4 | 4
  ADLs: Change at Month 114 | 5.6 (1.2) | -0.3 (1.2)
  ADLs: Change at Month 126: number analyzed (Participants) | 2 | 2
  ADLs: Change at Month 126 | 7.5 (1.6) | 1.5 (1.6)
  ADLs: Change at Month 138: number analyzed (Participants) | 1 | 1
  ADLs: Change at Month 138 | 12.8 (2.2) | 7.2 (2.2)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 6: number analyzed (Participants) | 38 | 36
  Physical Functioning/Large Fiber Neuropathy: Change at Month 6 | -2.3 (1.7) | -1.0 (1.7)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 12: number analyzed (Participants) | 38 | 36
  Physical Functioning/Large Fiber Neuropathy: Change at Month 12 | -2.9 (1.7) | 1.0 (1.7)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 18: number analyzed (Participants) | 38 | 36
  Physical Functioning/Large Fiber Neuropathy: Change at Month 18 | -2.7 (1.7) | 2.7 (1.7)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 24: number analyzed (Participants) | 38 | 36
  Physical Functioning/Large Fiber Neuropathy: Change at Month 24 | -3.2 (1.7) | -0.5 (1.7)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 30: number analyzed (Participants) | 37 | 36
  Physical Functioning/Large Fiber Neuropathy: Change at Month 30 | -1.0 (1.7) | 1.9 (1.7)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 42: number analyzed (Participants) | 36 | 33
  Physical Functioning/Large Fiber Neuropathy: Change at Month 42 | 0.6 (1.7) | -0.1 (1.8)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 54: number analyzed (Participants) | 36 | 33
  Physical Functioning/Large Fiber Neuropathy: Change at Month 54 | 0.8 (1.7) | -0.4 (1.8)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 66: number analyzed (Participants) | 33 | 31
  Physical Functioning/Large Fiber Neuropathy: Change at Month 66 | 1.3 (1.7) | 2.1 (1.8)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 78: number analyzed (Participants) | 9 | 6
  Physical Functioning/Large Fiber Neuropathy: Change at Month 78 | 2.6 (2.5) | -2.6 (2.9)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 90: number analyzed (Participants) | 7 | 5
  Physical Functioning/Large Fiber Neuropathy: Change at Month 90 | -0.7 (2.8) | 0.1 (3.2)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 102: number analyzed (Participants) | 5 | 4
  Physical Functioning/Large Fiber Neuropathy: Change at Month 102 | 7.0 (3.1) | -3.6 (3.5)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 114: number analyzed (Participants) | 4 | 4
  Physical Functioning/Large Fiber Neuropathy: Change at Month 114 | 7.2 (3.5) | -4.1 (3.5)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 126: number analyzed (Participants) | 2 | 2
  Physical Functioning/Large Fiber Neuropathy: Change at Month 126 | 24.8 (4.7) | 1.8 (4.7)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 138: number analyzed (Participants) | 1 | 1
  Physical Functioning/Large Fiber Neuropathy: Change at Month 138 | 24.7 (6.5) | 8.9 (6.5)
  Small Fiber Neuropathy: Change at Month 6: number analyzed (Participants) | 38 | 36
  Small Fiber Neuropathy: Change at Month 6 | 0.2 (0.5) | 0.5 (0.5)
  Small Fiber Neuropathy: Change at Month 12: number analyzed (Participants) | 38 | 36
  Small Fiber Neuropathy: Change at Month 12 | 0.5 (0.5) | 1.8 (0.5)
  Small Fiber Neuropathy: Change at Month 18: number analyzed (Participants) | 38 | 36
  Small Fiber Neuropathy: Change at Month 18 | 0.4 (0.5) | 1.5 (0.5)
  Small Fiber Neuropathy: Change at Month 24: number analyzed (Participants) | 38 | 36
  Small Fiber Neuropathy: Change at Month 24 | 0.3 (0.5) | 1.6 (0.5)
  Small Fiber Neuropathy: Change at Month 30: number analyzed (Participants) | 37 | 36
  Small Fiber Neuropathy: Change at Month 30 | 1.1 (0.5) | 2.0 (0.5)
  Small Fiber Neuropathy: Change at Month 42: number analyzed (Participants) | 36 | 33
  Small Fiber Neuropathy: Change at Month 42 | 1.7 (0.5) | 2.2 (0.5)
  Small Fiber Neuropathy: Change at Month 54: number analyzed (Participants) | 36 | 33
  Small Fiber Neuropathy: Change at Month 54 | 1.9 (0.5) | 1.6 (0.5)
  Small Fiber Neuropathy: Change at Month 66: number analyzed (Participants) | 33 | 31
  Small Fiber Neuropathy: Change at Month 66 | 1.9 (0.5) | 1.8 (0.5)
  Small Fiber Neuropathy: Change at Month 78: number analyzed (Participants) | 9 | 6
  Small Fiber Neuropathy: Change at Month 78 | 1.9 (0.8) | 1.3 (0.9)
  Small Fiber Neuropathy: Change at Month 90: number analyzed (Participants) | 7 | 5
  Small Fiber Neuropathy: Change at Month 90 | 1.7 (0.9) | 1.1 (1.0)
  Small Fiber Neuropathy: Change at Month 102: number analyzed (Participants) | 5 | 4
  Small Fiber Neuropathy: Change at Month 102 | 3.0 (1.0) | 1.2 (1.1)
  Small Fiber Neuropathy: Change at Month 114: number analyzed (Participants) | 4 | 4
  Small Fiber Neuropathy: Change at Month 114 | 2.8 (1.1) | 1.2 (1.1)
  Small Fiber Neuropathy: Change at Month 126: number analyzed (Participants) | 2 | 2
  Small Fiber Neuropathy: Change at Month 126 | 8.3 (1.4) | 1.1 (1.5)
  Small Fiber Neuropathy: Change at Month 138: number analyzed (Participants) | 1 | 1
  Small Fiber Neuropathy: Change at Month 138 | 11.8 (2.0) | 6.8 (2.0)
  Autonomic Neuropathy: Change at Month 6: number analyzed (Participants) | 38 | 36
  Autonomic Neuropathy: Change at Month 6 | -0.1 (0.3) | 0.0 (0.4)
  Autonomic Neuropathy: Change at Month 12: number analyzed (Participants) | 38 | 36
  Autonomic Neuropathy: Change at Month 12 | -0.3 (0.3) | 0.3 (0.4)
  Autonomic Neuropathy: Change at Month 18: number analyzed (Participants) | 38 | 36
  Autonomic Neuropathy: Change at Month 18 | 0.0 (0.3) | 0.5 (0.4)
  Autonomic Neuropathy: Change at Month 24: number analyzed (Participants) | 38 | 36
  Autonomic Neuropathy: Change at Month 24 | -0.2 (0.3) | 0.0 (0.4)
  Autonomic Neuropathy: Change at Month 30: number analyzed (Participants) | 37 | 36
  Autonomic Neuropathy: Change at Month 30 | 0.2 (0.3) | 0.2 (0.4)
  Autonomic Neuropathy: Change at Month 42: number analyzed (Participants) | 36 | 33
  Autonomic Neuropathy: Change at Month 42 | -0.3 (0.3) | -0.7 (0.4)
  Autonomic Neuropathy: Change at Month 54: number analyzed (Participants) | 36 | 33
  Autonomic Neuropathy: Change at Month 54 | -0.5 (0.3) | -0.4 (0.4)
  Autonomic Neuropathy: Change at Month 66: number analyzed (Participants) | 33 | 31
  Autonomic Neuropathy: Change at Month 66 | -0.3 (0.4) | -0.3 (0.4)
  Autonomic Neuropathy: Change at Month 78: number analyzed (Participants) | 9 | 6
  Autonomic Neuropathy: Change at Month 78 | 0.1 (0.6) | -1.1 (0.7)
  Autonomic Neuropathy: Change at Month 90: number analyzed (Participants) | 7 | 5
  Autonomic Neuropathy: Change at Month 90 | -0.6 (0.6) | -1.9 (0.7)
  Autonomic Neuropathy: Change at Month 102: number analyzed (Participants) | 5 | 4
  Autonomic Neuropathy: Change at Month 102 | 0.8 (0.7) | -1.4 (0.8)
  Autonomic Neuropathy: Change at Month 114: number analyzed (Participants) | 4 | 4
  Autonomic Neuropathy: Change at Month 114 | 1.2 (0.8) | -2.4 (0.8)
  Autonomic Neuropathy: Change at Month 126: number analyzed (Participants) | 2 | 2
  Autonomic Neuropathy: Change at Month 126 | 1.6 (1.1) | -1.2 (1.1)
  Autonomic Neuropathy: Change at Month 138: number analyzed (Participants) | 1 | 1
  Autonomic Neuropathy: Change at Month 138 | 1.9 (1.5) | -0.7 (1.5)

33. Secondary Outcome: NonVal30Met Group: Change From B3461022 Baseline in Total Quality of Life (TQOL) Score Assessed Using Norfolk Quality of Life for Diabetic Neuropathy (QOL-DN) Questionnaire at Month 6, 24, 36, 48, 72, 84, 96, 108, 120
Description: as for outcome 7
Time Frame: Baseline of B3461022 (Fx1A-201), Month 6, 24, 36, 48, 72, 84, 96, 108, 120
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale
  TQOL: Change at Month 6: number analyzed (Participants) | 17
  TQOL: Change at Month 6 | -4.0 (5.8)
  TQOL: Change at Month 24 | 4.0 (5.7)
  TQOL: Change at Month 36: number analyzed (Participants) | 12
  TQOL: Change at Month 36 | 15.8 (6.3)
  TQOL: Change at Month 48: number analyzed (Participants) | 9
  TQOL: Change at Month 48 | 15.5 (6.9)
  TQOL: Change at Month 72: number analyzed (Participants) | 3
  TQOL: Change at Month 72 | 16.2 (10.1)
  TQOL: Change at Month 84: number analyzed (Participants) | 2
  TQOL: Change at Month 84 | 9.5 (11.9)
  TQOL: Change at Month 96: number analyzed (Participants) | 2
  TQOL: Change at Month 96 | 11.5 (11.9)
  TQOL: Change at Month 108: number analyzed (Participants) | 2
  TQOL: Change at Month 108 | 22.0 (11.9)
  TQOL: Change at Month 120: number analyzed (Participants) | 2
  TQOL: Change at Month 120 | 28.5 (11.9)

34. Secondary Outcome: NonVal30Met Group: TQOL Subscale Scores: Symptom, ADLs, Physical Functioning/Large Fiber Neuropathy, Small Fiber Neuropathy, Autonomic Neuropathy Assessed Using Norfolk QOL-DN at Baseline
Description: as for outcome 31
Time Frame: Baseline of B3461022 (Fx1A-201)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale
  Symptom: Baseline | 10.3 (7.3)
  ADLs: Baseline | 8.4 (6.9)
  Physical Functioning/Large Fiber Neuropathy: Baseline | 28.7 (18.1)
  Small Fiber Neuropathy: Baseline | 4.5 (5.0)
  Autonomic Neuropathy: Baseline | 2.0 (2.1)

35. Secondary Outcome: NonVal30Met Group: Change From Baseline in TQOL Subscale Scores: Symptom, ADLs, Physical Functioning/Large Fiber Neuropathy, Small Fiber Neuropathy, Autonomic Neuropathy Assessed Using Norfolk QOL-DN at Month 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120
Description: as for outcome 31
Time Frame: Baseline of B3461022 (Fx1A-201), Month 6, 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale
  Symptom: Change at Month 6: number analyzed (Participants) | 17
  Symptom: Change at Month 6 | -0.8 (1.1)
  Symptom: Change at Month 12 | 0.0 (1.1)
  Symptom: Change at Month 24: number analyzed (Participants) | 16
  Symptom: Change at Month 24 | -0.1 (1.1)
  Symptom: Change at Month 36: number analyzed (Participants) | 10
  Symptom: Change at Month 36 | 2.9 (1.3)
  Symptom: Change at Month 48: number analyzed (Participants) | 9
  Symptom: Change at Month 48 | 4.1 (1.3)
  Symptom: Change at Month 60: number analyzed (Participants) | 7
  Symptom: Change at Month 60 | 2.6 (1.4)
  Symptom: Change at Month 72: number analyzed (Participants) | 3
  Symptom: Change at Month 72 | 2.5 (1.9)
  Symptom: Change at Month 84: number analyzed (Participants) | 2
  Symptom: Change at Month 84 | 0.5 (2.3)
  Symptom: Change at Month 96: number analyzed (Participants) | 2
  Symptom: Change at Month 96 | 1.0 (2.3)
  Symptom: Change at Month 108: number analyzed (Participants) | 2
  Symptom: Change at Month 108 | 2.5 (2.3)
  Symptom: Change at Month 120: number analyzed (Participants) | 2
  Symptom: Change at Month 120 | -0.5 (2.3)
  ADLs: Change at Month 6: number analyzed (Participants) | 17
  ADLs: Change at Month 6 | 0.1 (1.1)
  ADLs: Change at Month 12 | 1.1 (1.1)
  ADLs: Change at Month 24 | 1.8 (1.1)
  ADLs: Change at Month 36: number analyzed (Participants) | 12
  ADLs: Change at Month 36 | 3.5 (1.2)
  ADLs: Change at Month 48: number analyzed (Participants) | 9
  ADLs: Change at Month 48 | 3.5 (1.3)
  ADLs: Change at Month 60: number analyzed (Participants) | 7
  ADLs: Change at Month 60 | 3.1 (1.4)
  ADLs: Change at Month 72: number analyzed (Participants) | 3
  ADLs: Change at Month 72 | 3.4 (1.9)
  ADLs: Change at Month 84: number analyzed (Participants) | 2
  ADLs: Change at Month 84 | 3.2 (2.3)
  ADLs: Change at Month 96: number analyzed (Participants) | 2
  ADLs: Change at Month 96 | 3.2 (2.3)
  ADLs: Change at Month 108: number analyzed (Participants) | 2
  ADLs: Change at Month 108 | 4.2 (2.3)
  ADLs: Change at Month 120: number analyzed (Participants) | 2
  ADLs: Change at Month 120 | 8.2 (2.3)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 6: number analyzed (Participants) | 17
  Physical Functioning/Large Fiber Neuropathy: Change at Month 6 | -2.1 (3.4)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 12 | -0.6 (3.3)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 24 | 0.6 (3.3)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 36: number analyzed (Participants) | 12
  Physical Functioning/Large Fiber Neuropathy: Change at Month 36 | 7.1 (3.7)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 48: number analyzed (Participants) | 9
  Physical Functioning/Large Fiber Neuropathy: Change at Month 48 | 5.8 (4.0)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 60: number analyzed (Participants) | 7
  Physical Functioning/Large Fiber Neuropathy: Change at Month 60 | 5.5 (4.3)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 72: number analyzed (Participants) | 3
  Physical Functioning/Large Fiber Neuropathy: Change at Month 72 | 4.5 (5.8)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 84: number analyzed (Participants) | 2
  Physical Functioning/Large Fiber Neuropathy: Change at Month 84 | 2.9 (6.8)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 96: number analyzed (Participants) | 2
  Physical Functioning/Large Fiber Neuropathy: Change at Month 96 | 5.4 (6.8)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 108: number analyzed (Participants) | 2
  Physical Functioning/Large Fiber Neuropathy: Change at Month 108 | 11.4 (6.8)
  Physical Functioning/Large Fiber Neuropathy: Change at Month 120: number analyzed (Participants) | 2
  Physical Functioning/Large Fiber Neuropathy: Change at Month 120 | 15.4 (6.8)
  Small Fiber Neuropathy: Change at Month 6: number analyzed (Participants) | 17
  Small Fiber Neuropathy: Change at Month 6 | -0.4 (0.9)
  Small Fiber Neuropathy: Change at Month 12 | 0.9 (0.9)
  Small Fiber Neuropathy: Change at Month 24 | 0.9 (0.9)
  Small Fiber Neuropathy: Change at Month 36: number analyzed (Participants) | 12
  Small Fiber Neuropathy: Change at Month 36 | 1.6 (1.0)
  Small Fiber Neuropathy: Change at Month 48: number analyzed (Participants) | 9
  Small Fiber Neuropathy: Change at Month 48 | 2.2 (1.2)
  Small Fiber Neuropathy: Change at Month 60: number analyzed (Participants) | 7
  Small Fiber Neuropathy: Change at Month 60 | 1.5 (1.3)
  Small Fiber Neuropathy: Change at Month 72: number analyzed (Participants) | 3
  Small Fiber Neuropathy: Change at Month 72 | 4.1 (1.7)
  Small Fiber Neuropathy: Change at Month 84: number analyzed (Participants) | 2
  Small Fiber Neuropathy: Change at Month 84 | 2.1 (2.1)
  Small Fiber Neuropathy: Change at Month 96: number analyzed (Participants) | 2
  Small Fiber Neuropathy: Change at Month 96 | 1.6 (2.1)
  Small Fiber Neuropathy: Change at Month 108: number analyzed (Participants) | 2
  Small Fiber Neuropathy: Change at Month 108 | 2.6 (2.1)
  Small Fiber Neuropathy: Change at Month 120: number analyzed (Participants) | 2
  Small Fiber Neuropathy: Change at Month 120 | 2.1 (2.1)
  Autonomic Neuropathy: Change at Month 6: number analyzed (Participants) | 17
  Autonomic Neuropathy: Change at Month 6 | -0.5 (0.4)
  Autonomic Neuropathy: Change at Month 12 | 0.0 (0.4)
  Autonomic Neuropathy: Change at Month 24 | 0.2 (0.4)
  Autonomic Neuropathy: Change at Month 36: number analyzed (Participants) | 12
  Autonomic Neuropathy: Change at Month 36 | 0.1 (0.4)
  Autonomic Neuropathy: Change at Month 48: number analyzed (Participants) | 9
  Autonomic Neuropathy: Change at Month 48 | 0.3 (0.5)
  Autonomic Neuropathy: Change at Month 60: number analyzed (Participants) | 7
  Autonomic Neuropathy: Change at Month 60 | 0.2 (0.6)
  Autonomic Neuropathy: Change at Month 72: number analyzed (Participants) | 3
  Autonomic Neuropathy: Change at Month 72 | 1.6 (0.8)
  Autonomic Neuropathy: Change at Month 84: number analyzed (Participants) | 2
  Autonomic Neuropathy: Change at Month 84 | 0.6 (1.0)
  Autonomic Neuropathy: Change at Month 96: number analyzed (Participants) | 2
  Autonomic Neuropathy: Change at Month 96 | 0.1 (1.0)
  Autonomic Neuropathy: Change at Month 108: number analyzed (Participants) | 2
  Autonomic Neuropathy: Change at Month 108 | 1.1 (1.0)
  Autonomic Neuropathy: Change at Month 120: number analyzed (Participants) | 2
  Autonomic Neuropathy: Change at Month 120 | 3.1 (1.0)

36. Secondary Outcome: Val30Met Group: Karnofsky Performance Scale (KPS) Score at Month 42, 54, 78, 90, 102, 114, 126 and 138
Description: as for outcome 15
Time Frame: Baseline of B3461023, Month 42, 54, 78, 90, 102, 114, 126 and 138
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
units on a scale
  Month 42: number analyzed (Participants) | 37 | 34
  Month 42 | 83.8 (11.63) | 81.5 (11.32)
  Month 54: number analyzed (Participants) | 36 | 34
  Month 54 | 86.1 (10.22) | 82.1 (11.49)
  Month 78: number analyzed (Participants) | 9 | 7
  Month 78 | 78.9 (14.53) | 81.4 (16.76)
  Month 90: number analyzed (Participants) | 9 | 6
  Month 90 | 75.6 (15.09) | 81.7 (14.72)
  Month 102: number analyzed (Participants) | 7 | 5
  Month 102 | 68.6 (16.76) | 80.0 (10.00)
  Month 114: number analyzed (Participants) | 4 | 4
  Month 114 | 75.0 (12.91) | 82.5 (9.57)
  Month 126: number analyzed (Participants) | 2 | 2
  Month 126 | 75.0 (7.07) | 75.0 (21.21)
  Month 138: number analyzed (Participants) | 1 | 1
  Month 138 | 70.0 (NA) — The upper limit of 95% CI could not be estimated due to less number of participants with event. | 60.0 (NA) — The upper limit of 95% CI could not be estimated due to less number of participants with event.

37. Secondary Outcome: NonVal30Met Group: Change From B3461022 Baseline in Karnofsky Performance Scale (KPS) Score at Month 6, 24, 36, 48, 72, 84, 96, 108 and 120
Description: as for outcome 15
Time Frame: Baseline of B3461022, Month 6, 24, 36, 48, 72, 84, 96, 108 and 120
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
units on a scale
  Change at Month 6 | -0.9 (2.57)
  Change at Month 24 | -5.3 (2.57)
  Change at Month 36: number analyzed (Participants) | 11
  Change at Month 36 | -4.8 (3.09)
  Change at Month 48: number analyzed (Participants) | 10
  Change at Month 48 | -10.6 (3.22)
  Change at Month 72: number analyzed (Participants) | 4
  Change at Month 72 | -10.1 (4.76)
  Change at Month 84: number analyzed (Participants) | 2
  Change at Month 84 | -3.3 (6.56)
  Change at Month 96: number analyzed (Participants) | 2
  Change at Month 96 | -3.3 (6.56)
  Change at Month 108: number analyzed (Participants) | 2
  Change at Month 108 | -3.3 (6.56)
  Change at Month 120: number analyzed (Participants) | 2
  Change at Month 120 | -33.3 (6.56)

38. Secondary Outcome: Val30Met Group: Number of Participants by Ambulation Stage at Week 12, Month 6, 9, 12, 18, 21, 24, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 69, 72, 75, 78, 81, 84, 87, 90, 93, 96, 99, 102, 105, 108, 111, 114, 117, 120, 123, 126, 129
Description: as for outcome 19
Time Frame: Week 12, Month 6, 9, 12, 18, 21, 24, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78, 81, 84, 87, 90, 93, 96, 99, 102, 105, 108, 111, 114, 117, 120, 123, 126 and 129
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis
Number analyzed (Participants) | 38 | 37
Participants
  Week 12: number analyzed (Participants) | 37 | 36
  Week 12: Stage 1 (Normal) | 37 | 36
  Week 12: Stage 2 (Some assistance required) | 0 | 0
  Week 12: Stage 3 (Not ambulatory) | 0 | 0
  Month 6: number analyzed (Participants) | 37 | 36
  Month 6: Stage 1 (Normal) | 37 | 36
  Month 6: Stage 2 (Some assistance required) | 0 | 0
  Month 6: Stage 3 (Not ambulatory) | 0 | 0
  Month 9: number analyzed (Participants) | 37 | 36
  Month 9: Stage 1 (Normal) | 37 | 36
  Month 9: Stage 2 (Some assistance required) | 0 | 0
  Month 9: Stage 3 (Not ambulatory) | 0 | 0
  Month 12: number analyzed (Participants) | 37 | 36
  Month 12: Stage 1 (Normal) | 37 | 36
  Month 12: Stage 2 (Some assistance required) | 0 | 0
  Month 12: Stage 3 (Not ambulatory) | 0 | 0
  Month 18: number analyzed (Participants) | 37 | 36
  Month 18: Stage 1 (Normal) | 37 | 36
  Month 18: Stage 2 (Some assistance required) | 0 | 0
  Month 18: Stage 3 (Not ambulatory) | 0 | 0
  Month 21: number analyzed (Participants) | 37 | 36
  Month 21: Stage 1 (Normal) | 37 | 36
  Month 21: Stage 2 (Some assistance required) | 0 | 0
  Month 21: Stage 3 (Not ambulatory) | 0 | 0
  Month 24: number analyzed (Participants) | 38 | 36
  Month 24: Stage 1 (Normal) | 37 | 36
  Month 24: Stage 2 (Some assistance required) | 0 | 0
  Month 24: Stage 3 (Not ambulatory) | 1 | 0
  Month 33: number analyzed (Participants) | 37 | 35
  Month 33: Stage 1 (Normal) | 37 | 34
  Month 33: Stage 2 (Some assistance required) | 0 | 1
  Month 33: Stage 3 (Not ambulatory) | 0 | 0
  Month 36: number analyzed (Participants) | 37 | 35
  Month 36: Stage 1 (Normal) | 35 | 34
  Month 36: Stage 2 (Some assistance required) | 2 | 1
  Month 36: Stage 3 (Not ambulatory) | 0 | 0
  Month 39: number analyzed (Participants) | 37 | 35
  Month 39: Stage 1 (Normal) | 35 | 34
  Month 39: Stage 2 (Some assistance required) | 2 | 1
  Month 39: Stage 3 (Not ambulatory) | 0 | 0
  Month 42: number analyzed (Participants) | 37 | 34
  Month 42: Stage 1 (Normal) | 36 | 33
  Month 42: Stage 2 (Some assistance required) | 1 | 1
  Month 42: Stage 3 (Not ambulatory) | 0 | 0
  Month 45: number analyzed (Participants) | 37 | 34
  Month 45: Stage 1 (Normal) | 36 | 33
  Month 45: Stage 2 (Some assistance required) | 1 | 1
  Month 45: Stage 3 (Not ambulatory) | 0 | 0
  Month 48: number analyzed (Participants) | 36 | 34
  Month 48: Stage 1 (Normal) | 34 | 32
  Month 48: Stage 2 (Some assistance required) | 2 | 2
  Month 48: Stage 3 (Not ambulatory) | 0 | 0
  Month 51: number analyzed (Participants) | 36 | 34
  Month 51: Stage 1 (Normal) | 34 | 31
  Month 51: Stage 2 (Some assistance required) | 2 | 3
  Month 51: Stage 3 (Not ambulatory) | 0 | 0
  Month 54: number analyzed (Participants) | 34 | 31
  Month 54: Stage 1 (Normal) | 32 | 27
  Month 54: Stage 2 (Some assistance required) | 2 | 4
  Month 54: Stage 3 (Not ambulatory) | 0 | 0
  Month 57: number analyzed (Participants) | 34 | 31
  Month 57: Stage 1 (Normal) | 32 | 27
  Month 57: Stage 2 (Some assistance required) | 2 | 4
  Month 57: Stage 3 (Not ambulatory) | 0 | 0
  Month 60: number analyzed (Participants) | 32 | 31
  Month 60: Stage 1 (Normal) | 30 | 26
  Month 60: Stage 2 (Some assistance required) | 2 | 5
  Month 60: Stage 3 (Not ambulatory) | 0 | 0
  Month 63: number analyzed (Participants) | 29 | 27
  Month 63: Stage 1 (Normal) | 27 | 22
  Month 63: Stage 2 (Some assistance required) | 2 | 5
  Month 63: Stage 3 (Not ambulatory) | 0 | 0
  Month 69: number analyzed (Participants) | 11 | 8
  Month 69: Stage 1 (Normal) | 9 | 5
  Month 69: Stage 2 (Some assistance required) | 2 | 3
  Month 69: Stage 3 (Not ambulatory) | 0 | 0
  Month 72: number analyzed (Participants) | 9 | 7
  Month 72: Stage 1 (Normal) | 8 | 5
  Month 72: Stage 2 (Some assistance required) | 1 | 2
  Month 72: Stage 3 (Not ambulatory) | 0 | 0
  Month 75: number analyzed (Participants) | 9 | 6
  Month 75: Stage 1 (Normal) | 8 | 4
  Month 75: Stage 2 (Some assistance required) | 1 | 2
  Month 75: Stage 3 (Not ambulatory) | 0 | 0
  Month 78: number analyzed (Participants) | 9 | 6
  Month 78: Stage 1 (Normal) | 8 | 4
  Month 78: Stage 2 (Some assistance required) | 1 | 2
  Month 78: Stage 3 (Not ambulatory) | 0 | 0
  Month 81: number analyzed (Participants) | 9 | 6
  Month 81: Stage 1 (Normal) | 8 | 4
  Month 81: Stage 2 (Some assistance required) | 1 | 2
  Month 81: Stage 3 (Not ambulatory) | 0 | 0
  Month 84: number analyzed (Participants) | 9 | 6
  Month 84: Stage 1 (Normal) | 8 | 4
  Month 84: Stage 2 (Some assistance required) | 1 | 2
  Month 84: Stage 3 (Not ambulatory) | 0 | 0
  Month 87: number analyzed (Participants) | 9 | 6
  Month 87: Stage 1 (Normal) | 8 | 4
  Month 87: Stage 2 (Some assistance required) | 1 | 2
  Month 87: Stage 3 (Not ambulatory) | 0 | 0
  Month 90: number analyzed (Participants) | 9 | 5
  Month 90: Stage 1 (Normal) | 7 | 3
  Month 90: Stage 2 (Some assistance required) | 2 | 2
  Month 90: Stage 3 (Not ambulatory) | 0 | 0
  Month 93: number analyzed (Participants) | 7 | 5
  Month 93: Stage 1 (Normal) | 5 | 3
  Month 93: Stage 2 (Some assistance required) | 2 | 2
  Month 93: Stage 3 (Not ambulatory) | 0 | 0
  Month 96: number analyzed (Participants) | 7 | 4
  Month 96: Stage 1 (Normal) | 5 | 3
  Month 96: Stage 2 (Some assistance required) | 1 | 1
  Month 96: Stage 3 (Not ambulatory) | 1 | 0
  Month 99: number analyzed (Participants) | 5 | 4
  Month 99: Stage 1 (Normal) | 4 | 3
  Month 99: Stage 2 (Some assistance required) | 1 | 1
  Month 99: Stage 3 (Not ambulatory) | 0 | 0
  Month 102: number analyzed (Participants) | 4 | 4
  Month 102: Stage 1 (Normal) | 3 | 3
  Month 102: Stage 2 (Some assistance required) | 1 | 1
  Month 102: Stage 3 (Not ambulatory) | 0 | 0
  Month 105: number analyzed (Participants) | 4 | 4
  Month 105: Stage 1 (Normal) | 3 | 3
  Month 105: Stage 2 (Some assistance required) | 1 | 1
  Month 105: Stage 3 (Not ambulatory) | 0 | 0
  Month 108: number analyzed (Participants) | 3 | 4
  Month 108: Stage 1 (Normal) | 2 | 3
  Month 108: Stage 2 (Some assistance required) | 1 | 1
  Month 108: Stage 3 (Not ambulatory) | 0 | 0
  Month 111: number analyzed (Participants) | 2 | 2
  Month 111: Stage 1 (Normal) | 2 | 1
  Month 111: Stage 2 (Some assistance required) | 0 | 1
  Month 111: Stage 3 (Not ambulatory) | 0 | 0
  Month 114: number analyzed (Participants) | 2 | 2
  Month 114: Stage 1 (Normal) | 2 | 1
  Month 114: Stage 2 (Some assistance required) | 0 | 1
  Month 114: Stage 3 (Not ambulatory) | 0 | 0
  Month 117: number analyzed (Participants) | 2 | 2
  Month 117: Stage 1 (Normal) | 2 | 1
  Month 117: Stage 2 (Some assistance required) | 0 | 1
  Month 117: Stage 3 (Not ambulatory) | 0 | 0
  Month 120: number analyzed (Participants) | 2 | 2
  Month 120: Stage 1 (Normal) | 2 | 1
  Month 120: Stage 2 (Some assistance required) | 0 | 1
  Month 120: Stage 3 (Not ambulatory) | 0 | 0
  Month 123: number analyzed (Participants) | 2 | 2
  Month 123: Stage 1 (Normal) | 2 | 1
  Month 123: Stage 2 (Some assistance required) | 0 | 1
  Month 123: Stage 3 (Not ambulatory) | 0 | 0
  Month 126: number analyzed (Participants) | 2 | 2
  Month 126: Stage 1 (Normal) | 2 | 1
  Month 126: Stage 2 (Some assistance required) | 0 | 1
  Month 126: Stage 3 (Not ambulatory) | 0 | 0
  Month 129: number analyzed (Participants) | 1 | 1
  Month 129: Stage 1 (Normal) | 1 | 0
  Month 129: Stage 2 (Some assistance required) | 0 | 1
  Month 129: Stage 3 (Not ambulatory) | 0 | 0

39. Secondary Outcome: NonVal30Met Group: Number of Participants by Ambulation Stage at Month 3, 6, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 63, 66, 69, 72, 75, 78, 81, 84, 87, 90, 93, 96, 99, 102, 105, 108, 111, 114, 117, 120, 123, 126, 129
Description: as for outcome 21
Time Frame: Month 3, 6, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 63, 66, 69, 72, 75, 78, 81, 84, 87, 90, 93, 96, 99, 102, 105, 108, 111, 114, 117, 120, 123, 126 and 129
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | NonVal30Met: Tafamidis
Number analyzed (Participants) | 18
Participants
  Month 3: number analyzed (Participants) | 12
  Month 3: Stage 1 (Normal) | 7
  Month 3: Stage 2 (Some assistance required) | 5
  Month 3: Stage 3 (Not ambulatory) | 0
  Month 6: number analyzed (Participants) | 12
  Month 6: Stage 1 (Normal) | 7
  Month 6: Stage 2 (Some assistance required) | 5
  Month 6: Stage 3 (Not ambulatory) | 0
  Month 15: number analyzed (Participants) | 14
  Month 15: Stage 1 (Normal) | 7
  Month 15: Stage 2 (Some assistance required) | 5
  Month 15: Stage 3 (Not ambulatory) | 2
  Month 18: number analyzed (Participants) | 15
  Month 18: Stage 1 (Normal) | 7
  Month 18: Stage 2 (Some assistance required) | 6
  Month 18: Stage 3 (Not ambulatory) | 2
  Month 21: number analyzed (Participants) | 15
  Month 21: Stage 1 (Normal) | 7
  Month 21: Stage 2 (Some assistance required) | 6
  Month 21: Stage 3 (Not ambulatory) | 2
  Month 24: number analyzed (Participants) | 16
  Month 24: Stage 1 (Normal) | 8
  Month 24: Stage 2 (Some assistance required) | 6
  Month 24: Stage 3 (Not ambulatory) | 2
  Month 27: number analyzed (Participants) | 15
  Month 27: Stage 1 (Normal) | 7
  Month 27: Stage 2 (Some assistance required) | 7
  Month 27: Stage 3 (Not ambulatory) | 1
  Month 30: number analyzed (Participants) | 13
  Month 30: Stage 1 (Normal) | 5
  Month 30: Stage 2 (Some assistance required) | 7
  Month 30: Stage 3 (Not ambulatory) | 1
  Month 33: number analyzed (Participants) | 13
  Month 33: Stage 1 (Normal) | 4
  Month 33: Stage 2 (Some assistance required) | 8
  Month 33: Stage 3 (Not ambulatory) | 1
  Month 36: number analyzed (Participants) | 13
  Month 36: Stage 1 (Normal) | 3
  Month 36: Stage 2 (Some assistance required) | 9
  Month 36: Stage 3 (Not ambulatory) | 1
  Month 39: number analyzed (Participants) | 12
  Month 39: Stage 1 (Normal) | 3
  Month 39: Stage 2 (Some assistance required) | 8
  Month 39: Stage 3 (Not ambulatory) | 1
  Month 42: number analyzed (Participants) | 10
  Month 42: Stage 1 (Normal) | 2
  Month 42: Stage 2 (Some assistance required) | 6
  Month 42: Stage 3 (Not ambulatory) | 2
  Month 45: number analyzed (Participants) | 8
  Month 45: Stage 1 (Normal) | 1
  Month 45: Stage 2 (Some assistance required) | 6
  Month 45: Stage 3 (Not ambulatory) | 1
  Month 48: number analyzed (Participants) | 7
  Month 48: Stage 1 (Normal) | 2
  Month 48: Stage 2 (Some assistance required) | 5
  Month 48: Stage 3 (Not ambulatory) | 0
  Month 51: number analyzed (Participants) | 7
  Month 51: Stage 1 (Normal) | 1
  Month 51: Stage 2 (Some assistance required) | 6
  Month 51: Stage 3 (Not ambulatory) | 0
  Month 54: number analyzed (Participants) | 7
  Month 54: Stage 1 (Normal) | 1
  Month 54: Stage 2 (Some assistance required) | 6
  Month 54: Stage 3 (Not ambulatory) | 0
  Month 57: number analyzed (Participants) | 7
  Month 57: Stage 1 (Normal) | 1
  Month 57: Stage 2 (Some assistance required) | 6
  Month 57: Stage 3 (Not ambulatory) | 0
  Month 63: number analyzed (Participants) | 4
  Month 63: Stage 1 (Normal) | 1
  Month 63: Stage 2 (Some assistance required) | 3
  Month 63: Stage 3 (Not ambulatory) | 0
  Month 66: number analyzed (Participants) | 4
  Month 66: Stage 1 (Normal) | 1
  Month 66: Stage 2 (Some assistance required) | 3
  Month 66: Stage 3 (Not ambulatory) | 0
  Month 69: number analyzed (Participants) | 3
  Month 69: Stage 1 (Normal) | 1
  Month 69: Stage 2 (Some assistance required) | 2
  Month 69: Stage 3 (Not ambulatory) | 0
  Month 72: number analyzed (Participants) | 3
  Month 72: Stage 1 (Normal) | 1
  Month 72: Stage 2 (Some assistance required) | 2
  Month 72: Stage 3 (Not ambulatory) | 0
  Month 75: number analyzed (Participants) | 2
  Month 75: Stage 1 (Normal) | 1
  Month 75: Stage 2 (Some assistance required) | 1
  Month 75: Stage 3 (Not ambulatory) | 0
  Month 78: number analyzed (Participants) | 2
  Month 78: Stage 1 (Normal) | 1
  Month 78: Stage 2 (Some assistance required) | 1
  Month 78: Stage 3 (Not ambulatory) | 0
  Month 81: number analyzed (Participants) | 2
  Month 81: Stage 1 (Normal) | 1
  Month 81: Stage 2 (Some assistance required) | 1
  Month 81: Stage 3 (Not ambulatory) | 0
  Month 84: number analyzed (Participants) | 2
  Month 84: Stage 1 (Normal) | 1
  Month 84: Stage 2 (Some assistance required) | 1
  Month 84: Stage 3 (Not ambulatory) | 0
  Month 87: number analyzed (Participants) | 2
  Month 87: Stage 1 (Normal) | 1
  Month 87: Stage 2 (Some assistance required) | 1
  Month 87: Stage 3 (Not ambulatory) | 0
  Month 90: number analyzed (Participants) | 2
  Month 90: Stage 1 (Normal) | 1
  Month 90: Stage 2 (Some assistance required) | 1
  Month 90: Stage 3 (Not ambulatory) | 0
  Month 93: number analyzed (Participants) | 2
  Month 93: Stage 1 (Normal) | 1
  Month 93: Stage 2 (Some assistance required) | 1
  Month 93: Stage 3 (Not ambulatory) | 0
  Month 96: number analyzed (Participants) | 2
  Month 96: Stage 1 (Normal) | 1
  Month 96: Stage 2 (Some assistance required) | 1
  Month 96: Stage 3 (Not ambulatory) | 0
  Month 99: number analyzed (Participants) | 2
  Month 99: Stage 1 (Normal) | 1
  Month 99: Stage 2 (Some assistance required) | 1
  Month 99: Stage 3 (Not ambulatory) | 0
  Month 102: number analyzed (Participants) | 2
  Month 102: Stage 1 (Normal) | 1
  Month 102: Stage 2 (Some assistance required) | 1
  Month 102: Stage 3 (Not ambulatory) | 0
  Month 105: number analyzed (Participants) | 2
  Month 105: Stage 1 (Normal) | 1
  Month 105: Stage 2 (Some assistance required) | 1
  Month 105: Stage 3 (Not ambulatory) | 0
  Month 108: number analyzed (Participants) | 2
  Month 108: Stage 1 (Normal) | 1
  Month 108: Stage 2 (Some assistance required) | 1
  Month 108: Stage 3 (Not ambulatory) | 0
  Month 111: number analyzed (Participants) | 2
  Month 111: Stage 1 (Normal) | 1
  Month 111: Stage 2 (Some assistance required) | 1
  Month 111: Stage 3 (Not ambulatory) | 0
  Month 114: number analyzed (Participants) | 2
  Month 114: Stage 1 (Normal) | 1
  Month 114: Stage 2 (Some assistance required) | 1
  Month 114: Stage 3 (Not ambulatory) | 0
  Month 117: number analyzed (Participants) | 2
  Month 117: Stage 1 (Normal) | 1
  Month 117: Stage 2 (Some assistance required) | 1
  Month 117: Stage 3 (Not ambulatory) | 0
  Month 120: number analyzed (Participants) | 2
  Month 120: Stage 1 (Normal) | 1
  Month 120: Stage 2 (Some assistance required) | 1
  Month 120: Stage 3 (Not ambulatory) | 0
  Month 123: number analyzed (Participants) | 2
  Month 123: Stage 1 (Normal) | 1
  Month 123: Stage 2 (Some assistance required) | 1
  Month 123: Stage 3 (Not ambulatory) | 0
  Month 126: number analyzed (Participants) | 1
  Month 126: Stage 1 (Normal) | 1
  Month 126: Stage 2 (Some assistance required) | 0
  Month 126: Stage 3 (Not ambulatory) | 0
  Month 129: number analyzed (Participants) | 1
  Month 129: Stage 1 (Normal) | 1
  Month 129: Stage 2 (Some assistance required) | 0
  Month 129: Stage 3 (Not ambulatory) | 0

40. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious AEs
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent AEs were events that emerged after enrollment in B3461023 (Fx1A-303) or which worsened during the course of B3461023 (Fx1A-303) relative to the pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: From Baseline (i.e., Day 0 of B3461023) up to 10 years
Population: Safety population included all enrolled participants in the current study B3461023 (Fx1A-303) and who had taken at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis
Number analyzed (Participants) | 38 | 37 | 18
Participants
  Treatment-Emergent AEs | 35 | 33 | 18
  Treatment-emergent SAEs | 6 | 9 | 10

41. Secondary Outcome: Number of Participants With Abnormality in Physical Examinations
Description: Complete physical examination included examination of the general appearance, head and neck, ears, eyes, nose, throat, respiratory, genitourinary, endocrine, cardiovascular, abdomen, skin, musculoskeletal, neurological, immunologic/allergies, hematologic/lymphatic. Abnormality in physical findings were based on investigator's decision.
Time Frame: From Baseline (i.e., Day 0 of B3461023) up to 10 years
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis
Number analyzed (Participants) | 38 | 37 | 18
Participants | 29 | 32 | 14

42. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Abnormalities criteria: Serum chemistry (bilirubin>1.5*upper limit normal [ULN]; aspartate aminotransferase; alanine aminotransferase; alkaline phosphatase; gamma glutamyl transferase >3.0*ULN; albumin<0.8*lower limit normal [LLN],>1.2*ULN; blood urea nitrogen, creatinine>1.3*ULN; free T4, thyrotropin, thyroxine <0.8*LLN,>1.2*ULN; glucose<0.6*LLN,>1.5*ULN); Coagulation (prothrombin time, prothrombin int. normalized ratio >1.1*ULN); Hematology(basophils; eosinophils, monocytes >1.2*ULN; leukocytes <0.6*LLN,>1.5*ULN; lymphocytes, neutrophils <0.8*LLN, >1.2*ULN).
Time Frame: From Baseline (i.e., Day 0 of B3461023) up to 10 years
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis
Number analyzed (Participants) | 38 | 37 | 18
Participants | 21 | 21 | 12

43. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Twelve-lead ECGs were obtained for all participants. Criteria for QT interval, Bazett's correction formula (QTcB) and Fridericia's correction formula (QTcF): greater than (>) 450-480 millisecond (msec), >480-500 msec and >500 msec. Findings were considered to be abnormal based on investigator's decision.
Time Frame: From Baseline (i.e., Day 0 of B3461023) up to 10 years
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis
Number analyzed (Participants) | 38 | 37 | 18
Participants
  QT Interval (msec): >450-480 | 8 | 7 | 6
  QT Interval (msec): >480-500 | 3 | 2 | 4
  QT Interval (msec): >500 | 2 | 1 | 6
  Bazett's Correction Formula (QTcB) (msec): >450-480 | 14 | 20 | 11
  Bazett's Correction Formula (QTcB) (msec): >480-500 | 6 | 3 | 5
  Bazett's Correction Formula (QTcB) (msec): >500 | 5 | 3 | 5
  Fridericia's Correction Formula (QTcF) (msec): >450-480 | 7 | 7 | 7
  Fridericia's Correction Formula (QTcF) (msec): >480-500 | 4 | 2 | 3
  Fridericia's Correction Formula (QTcF) (msec): >500 | 5 | 3 | 5

44. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Criteria for clinically significant changes: Supine and standing systolic blood pressure (BP): decrease from baseline of less than or equal to (<=) -20 millimeter of mercury (mmHg), increase from baseline of greater than or equal to (>=) 20 mmHg, systolic BP <90 mmHg or >180 mmHg; Supine and standing diastolic BP: decrease from baseline of <=-15 mmHg, increase from baseline of >= 15 mmHg, diastolic BP <50 mmHg or >105 mmHg; Supine and standing pulse rate: decrease from baseline of <=-15 beats per minute (bpm), increase from baseline of >=15 bpm, pulse rate <50 bpm or >120 bpm; Weight: decrease from baseline of <=-7 percentage (%) or increase from baseline of >=7%.
Time Frame: From Baseline (i.e., Day 0 of B3461023) up to 10 years
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis
Number analyzed (Participants) | 38 | 37 | 18
Participants | 38 | 37 | 18

45. Secondary Outcome: Number of Participants With Any Concomitant Medications Usage
Description: Number of participants with any concomitant medications usage are reported.
Time Frame: From Baseline (i.e., Day 0 of B3461023) up to 10 years
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis
Number analyzed (Participants) | 38 | 37 | 18
Participants | 36 | 37 | 17

ADVERSE EVENTS:
Time Frame: From Baseline (i.e., Day 0 of B3461023) up to 10 years
Description: Same event may appear as both an AE and Serious Adverse Events (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Val30Met: Tafamidis Then Tafamidis | Val30Met: Placebo Then Tafamidis | NonVal30Met: Tafamidis
All-Cause Mortality (participants affected / at risk) | 3/38 | 1/37 | 7/18
Serious Adverse Events (participants affected / at risk) | 6/38 | 9/37 | 10/18
Other Adverse Events (participants affected / at risk) | 34/38 | 32/37 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Val30Met: Tafamidis Then Tafamidis (N=38) | Val30Met: Placebo Then Tafamidis (N=37) | NonVal30Met: Tafamidis (N=18)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Amyloidosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (4)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 2 (3)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Central Nervous System Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's Type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Transplant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Val30Met: Tafamidis Then Tafamidis (N=38) | Val30Met: Placebo Then Tafamidis (N=37) | NonVal30Met: Tafamidis (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Bundle Branch Block Bilateral (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Dry Eye (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Eye Pruritus (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 3 (3) | 1 (2)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 4 (6)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (4)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Early Satiety (General disorders) | 2 (2) | 0 (0) | 0 (0)
Exercise Tolerance Decreased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4) | 2 (2)
Gait Disturbance (General disorders) | 3 (3) | 1 (1) | 1 (1)
Implant Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema Peripheral (General disorders) | 3 (3) | 1 (2) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Burn Infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infected Skin Ulcer (Infections and infestations) | 4 (5) | 2 (3) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 7 (10) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (9) | 3 (3) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (4) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (3) | 2 (4)
Skin Infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 4 (6) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 3 (3) | 3 (4)
Urinary Tract Infection (Infections and infestations) | 6 (11) | 6 (10) | 2 (2)
Vaginal Infection (Infections and infestations) | 3 (6) | 2 (2) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Burns Second Degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 12 (25)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 3 (5) | 0 (0) | 0 (0)
Medication Error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 6 (10) | 5 (8) | 1 (1)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic Ulcer (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Blood Cholesterol Increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (4) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4) | 3 (4)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (10) | 2 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Balance Disorder (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Burning Sensation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 3 (4)
Fine Motor Skill Dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 4 (4) | 4 (5) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 1 (2) | 2 (2) | 5 (6)
Paraesthesia (Nervous system disorders) | 3 (5) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 3 (5) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 1 (1) | 2 (4)
Renal Failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 3 (6) | 2 (2) | 2 (2)
Walking Disability (Social circumstances) | 2 (2) | 4 (4) | 0 (0)
Carpal Tunnel Decompression (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (2) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 4 (4)
Peripheral Vascular Disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2012-06-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT00925002/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT00925002/SAP_001.pdf